Doc id 43CH1627 Clinical Study Protocol ♣ GALDERMA **MA-34970** 

Print date:

2023-04-18 09:24

A randomized, multi-center, evaluator-blinded, no-treatment controlled study to evaluate the effectiveness and safety of Restylane Defyne for correction of Chin Retrusion

Study product: Restylane Defyne

Clinical Trial Number (CTN): 43CH1627

Q-Med AB Sponsor:

Seminariegatan 21

SE-752 28 Uppsala, Sweden

Telephone: +46 18 474 90 00

Facsimile: +46 18 474 90 01

## **Confidentiality Statement**

This study protocol contains confidential information belonging to Q-Med AB. Except as may be otherwise agreed to in writing, by accepting or reviewing these materials, you agree to hold such information in confidence and neither disclose it to any third parties (except where required by applicable law) nor use it for any other purpose than in relation to the clinical study described herein.

Doc id

43CH1627 Clinical Study Protocol

**MA-34970** 

# Summary of Changes in Clinical Study Protocol 43CH1627 from Version 2.0 to Version 3.0

Added text is written in **bold** and deleted text is written as strikethrough.

| to the<br>n of the<br>se EC,<br>was deleted. | Group A: Up to 20 subjects (the first two eligible subjects per Treating Investigator, each site will have 2 Treating Investigators as maximum) will be enrolled as group A. These subjects will all receive treatment with Restylane Defyne. |
|---|---|
| | 1 |
| | Group B: Evaluator treatment-blinded group with aApproximately 148 subjects will be randomized in a 3:1 ratio to Treatment Group or no-treatment Control Group, i.e., 111 subjects assigned to the Treatment Group and 37 subjects assigned to the Control Group. |
| to the n of the re EC, was deleted. | This is a randomized, evaluator-blinded, no-treatment controlled study in subjects with Chin Retrusion. Subjects will be screened for eligibility within 21 days prior to Baseline. The first 2 eligible subjects for each Treating Investigator will receive treatment as Group A. Before start of enrolment into Group B the injection technique will be evaluated by the Sponsor's Medical Expert and the Treating Investigator. The evaluation will be performed when the subjects in Group A for each Treating Investigator have received their first treatment at the baseline visit. During the evaluation it will be ensured that an appropriate injection technique has been used. An evaluation form will be completed by the Treating Investigator and sent to Sponsor's Medical Expert for assessment. If treatments are found to be correctly performed, no further training is needed, there are no outstanding questions regarding the injection technique and no other corrective actions are identified the enrolment in Group B can start for that Treating Investigator. The evaluation and decision to proceed with enrolment in Group B will be documented in writing. Eligible Ssubjects in group B will be randomized either to the Treatment Group or the Control Group in a 3:1 ratio. Summaries of the results for Group A and B will be done separately in the study report. Treatment Each subject assigned to Group A or the Treatment Group |

Title
43CH1627 Clinical Study Protocol Doc id ♣ GALDERMA MA-34970

| | | Subjects assigned to the Control Group in Group B will not receive treatment at baseline but will return for routine follow-up for 18 months. At month 6 visit after randomization, subjects in Control Group will be offered a treatment and, at the following visit, an optional touch-up treatment. |
|---|---|---|
| | | Evaluation of effectiveness |
| | | Chin Retrusion will be assessed using a separate Four-Point GCRS with photo guides by the Treating Investigator at each visit; and by the Blinded Evaluator at screening, baseline, 3, 6, 9 and 12 months after last treatment—in Group A and Treatment Group, |
| | | CCI |
| Synopsis-<br>Duration of<br>treatment and<br>follow-up | According to the suggestion of the leading site EC, Group A was deleted. | The total duration for each subject will be approximately 14 months for Group A and Treatment Group, 20 months for Control Group. |
| Synopsis-<br>Statistical<br>Methods | According to the suggestion of the leading site EC, Group A was deleted. | All summaries will be done separately for Group A and B. For statistical inference, only Group B will be used. |
| 4.1 General<br>Outline | According to the suggestion of the leading site EC, Group A was deleted. And Clarification | This is a randomized, evaluator-blinded, no-treatment controlled study in subjects with Chin Retrusion. Subjects will be screened for eligibility within 21 days prior to Baseline. The first 2 eligible subjects for each Treating Investigator will receive treatment as Group A. Before start of enrolment into Group B the injection technique will be evaluated by the Sponsor's Medical Expert and the Treating Investigator. The evaluation will be performed when the subjects in Group A for each Treating Investigator have received their first treatment at the baseline visit. During the evaluation it will be ensured that an appropriate injection technique has been used. An evaluation form will be completed by the Treating Investigator and sent to Sponsor's Medical Expert for assessment. If treatments are found to be correctly performed, no further training is needed, there are no outstanding questions regarding the injection technique and no other corrective actions are identified the enrolment in Group B can start for that Treating Investigator. The evaluation and decision to proceed with enrolment in Group B will be documented in writing. Eligible Ssubjects in group B will be randomized either to the Treatment Group or the Control Group in a 3:1 ratio. |
| | | Summaries of the results for Group A and B will be done |

Title
43CH1627 Clinical Study Protocol Doc id ♣ GALDERMA MA-34970

| | | separately in the study report. |
|---|---|---|
| | | <u>Treatment</u> |
| | | Each subject assigned to Group A or the Treatment Group in Group B will receive an initial treatment on Day 1. |
| | | Subjects assigned to the Control Group in Group B will not receive treatment at baseline but will return for routine follow-up for 18 months. At month 6 visit after randomization, subjects in Control Group will be offered a treatment and, at the following visit, an optional touch-up treatment. |
| | | Evaluation of effectiveness |
| | | Chin Retrusion will be assessed using a separate Four-Point GCRS with photo guides by the Treating Investigator at each visit; and by the Blinded Evaluator at screening, baseline, 3, 6, 9 and 12 months after last treatment—in Group A and Treatment Group, |
| | | CCI |
| | | *Figure 1, the Flow chart was changed accordingly. |
| 4.2 Number of<br>Subjects | According to the suggestion of the leading site EC, Group A was deleted. | approximately <del>168-</del> <b>148</b> subjects will be enrolled. |
| 4.3 Duration<br>of Subject<br>Participation | According to the suggestion of the leading site EC, Group A was deleted. | The total duration for each subject will be approximately 14 months for Group A and Treatment Group, 20 months for Control Group. |
| 4.4.1<br>Randomizatio<br>n | According to the suggestion of the leading site EC, | Approximately 148 subjects in group B will be randomized in a 3:1 ratio to treatment with Restylane Defyne or to no treatment. |
| | Group A was deleted. | Each subject will be assigned a subject number as they arrive for the treatment visit. For group B, FR andomization will be assigned via the eCRF system. |
| 4.4.1<br>Randomizatio<br>n | In the study, subjects will be randomized in eCRF, no additional randomization log is needed. | At the time for randomization, the subject's initials, date of randomization, subject number, randomized treatment, and the signature of the Investigator must be documented in a randomization log. |
| 4.7 Schedule of events | According to the suggestion of the leading site EC, Group A was deleted. | Table 1. Schedule of Events for Group A and Treatment Group |

43CH1627 Clinical Study Protocol Doc id ♣ GALDERMA MA-34970

| 4.7 Schedule | Typo error correction | Table 2. |
|---|---|---|
| of events | | CCI |
| 4.8.1 Visits for<br>Treatment<br>Group | According to the suggestion of the leading site EC, Group A was deleted. | 4.8.1 Visits for <del>Group A and</del> Treatment Group |
| 5.4 Screening<br>and Subject<br>Numbers | According to the suggestion of the leading site EC, Group A was deleted. | When the Investigator has confirmed that all inclusion criteria and no exclusion criteria are met, each enrolled subject will be assigned a subject number by the eCRF-For group A, consisting of a capital letter A, the site number, then followed by a consecutive number starting with 001 at each site, e.g. A1001, A1002; for group B, consisting of the site number followed by a consecutive number starting with 001 at each site, e.g. 1001, 1002. |
| 7.2 Galderma<br>Chin Retrusion<br>Scale (GCRS) | According to the suggestion of the leading site EC, Group A was deleted. | The Blinded Evaluator will rate the subject's Chin Retrusion using the GCRS at screening, baseline, 3, 6, 9 and 12 months after last treatment in Group A and Treatment Group; |
| CCI | According to the suggestion of the leading site EC, Group A was deleted. | CCI |
| 8.2 Laboratory assessment | Indirect bilirubin=total bilirubin-direct bilirubin, and in some labs it is not listed, so indirect bilirubin was deleted. | • Serum chemistry: renal function tests (creatinine and BUN); and liver function tests (aspartate amino transferase (ASAT), alanine amino transferase (ALAT) total bilirubin, and direct bilirubin and indirect bilirubin). |
| 10.1 General | According to the suggestion of the leading site EC, Group A was deleted. | A comprehensive Statistical Analysis Plan (SAP) with detailed description of all statistical analyses will be written and finalized prior to database lock (DBL). All summaries will be done separately for Group A and B. For group A, only descriptive statistics will be used. |
| 10.2 Analysis<br>Populations | According to the suggestion of the leading site EC, Group A was deleted. | <ul> <li>Safety Includes all subjects in Group B who were<br/>treated with Restylane Defyne or<br/>randomized to no-treatment group.<br/>Subjects are analyzed based on the as<br/>treated principle.</li> </ul> |
| | | <ul> <li>Full Includes all subjects in Group B who were<br/>Analysis treated with Restylane Defyne or<br/>Set (FAS) randomized to no-treatment group.<br/>Subjects are analysed according to the<br/>randomisation assignment.</li> </ul> |

| | Title | Doc id |
|------------|----------------------------------|----------|
| ♣ GALDERMA | 43CH1627 Clinical Study Protocol | MA-34970 |

| Subject | Updates required: |
|-----------------|-------------------|
| information | Yes No |
| and informed | res 🖂 NO 📋 |
| consent form | |
| Electronic case | Updates required: |
| report form | Yes No |
| (eCRF) | |

Doc id 43CH1627 Clinical Study Protocol ♣ GALDERMA **MA-34970** 

Print date:

2023-04-18 09:24

# **Study Administrative Structure**

Q-Med AB **Sponsor** 

Seminariegatan 21

SE-752 28 Uppsala, Sweden

Telephone: +46 18 474 90 00 Facsimile: +46 18 474 90 01

PPD PPD **Medical Expert** Clinical Project Manager Study Statistician

Further details on all participating Investigators and the complete administrative structure of the study are found in the study files. Note that administrative changes are to be documented in the study files without requiring a clinical study protocol (CSP) amendment.



## **Sponsor Signatures**

The CSP is electronically signed in the document management system within the Q-Med AB quality management system by the representatives listed below.



Electronically signed in the document management system within Q-Med quality management system

Sponsor's Medical Expert, Q-Med AB

Electronically signed in the document management system within Q-Med quality management system

Clinical Project Manager, Q-Med AB

Electronically signed in the document management system within Q-Med quality management system

Study Statistician, Q-Med AB PPD

Electronically signed in the document management system within Q-Med quality management system

| • | 43CH1627 Clinical Study Protocol | Doc id |
|-------------------|----------------------------------------|----------|
| <b>⊶</b> GALDERMA | 10 000000 0000000000000000000000000000 | MA-34970 |

Print date:

2023-04-18 09:24

| Signed Agreement of the Clinical Study Protocol | | |
|---|---|---|
| CTN:<br>Title of the CSP: | 43CH1627 A randomized, multi-center, evaluator-l treatment controlled study to evaluate and safety of Restylane Defyne for corrections. | the effectiveness |
| the contents. The study protoco | nd understand the protocol specified abo<br>ol, the Clinical Trial Agreement and the a<br>gator Brochure for Restylane Defyne will | dditional |
| Principal Investigator | | |
| Printed name | Signature | Date |
| Study site | | |

Title
43CH1627 Clinical Study Protocol Doc id ♣ GALDERMA MA-34970

Print date:

2023-04-18 09:24

# **Synopsis**

| Title of study: | A randomized, multi-center, evaluator-blinded, no-treatment controlled study to evaluate the effectiveness and safety of Restylane Defyne for correction of Chin Retrusion |
|---|---|
| Clinical Trial Number: | 43CH1627 |
| Countries involved,<br>number of<br>sites/country, number<br>of subjects: | The study will be conducted at approximately 5 sites in China. Approximately 148 subjects will be randomized in a 3:1 ratio to Treatment Group or no-treatment Control Group, i.e., 111 subjects assigned to the Treatment Group and 37 subjects assigned to the Control Group. |
| Objectives: | To evaluate the effectiveness and safety of Restylane Defyne versus a notreatment control in the treatment of Chin Retrusion. |
| Endpoints: | Primary effectiveness endpoint: |
| | <ul> <li>Percentage of responders, defined by at least 1 point improvement from<br/>baseline on the Galderma Chin Retrusion Scale (GCRS), as measured by the<br/>Blinded Evaluator at 6 months (after last treatment in Treatment Group, and<br/>after randomization in Control Group).</li> </ul> |
| | Secondary effectiveness endpoints: |
| | <ul> <li>Percentage of responders, defined by at least 1 point improvement from baseline on the GCRS, as measured by the Blinded Evaluator at 3, 9 and 12 months after last treatment in Treatment Group, and at 3 months after randomization, as well as 3, 6, 9 and 12 months after the last treatment in Control Group.</li> <li>Percentage of responders, defined by at least 1 point improvement from baseline on the GCRS, as measured by the Treating Investigator at each follow up visit.</li> </ul> |
| | CCI |
| | Safety endpoints: |
| | <ul> <li>Incidence, intensity, duration, and onset of adverse events (AEs) collected<br/>throughout the study.</li> </ul> |
| Study Design: | This is a randomized, evaluator-blinded, no-treatment controlled study in |

Doc id 43CH1627 Clinical Study Protocol GALDERMA MA-34970

subjects with Chin Retrusion.

Subjects will be screened for eligibility within 21 days prior to Baseline. Eligible subjects will be randomized either to the Treatment Group or the Control Group in a 3:1 ratio.

Print date:

2023-04-18 09:24

#### **Treatment**

Each subject assigned to the Treatment Group will receive an initial treatment on Day 1. A touch-up treatment may be performed 4 weeks after the initial treatment if optimal chin augmentation has not been obtained. Optimal chin augmentation is defined as the best possible aesthetic result that can be obtained for an individual study participant, as agreed upon by the Treating Investigator and subject. At least one (≥1) grade improvement from baseline on the GCRS should be the treatment target.

Subjects assigned to the Control Group will not receive treatment at baseline but will return for routine follow-up. At month 6 visit after randomization, subjects in Control Group will be offered a treatment and, at the following visit, an optional touch-up treatment.

#### **Evaluation of effectiveness**

Chin Retrusion will be assessed using a separate Four-Point GCRS with photo guides by the Treating Investigator at each visit; and by the Blinded Evaluator at screening, baseline, 3, 6, 9 and 12 months after last treatment in Treatment Group, and at screening, baseline, 3 and 6 months after randomization, as well as 3, 6, 9 and 12 months after last treatment in Control Group.



## Inclusion criteria:

The subject must meet the following criteria to be eligible for the study:

- 1. Signed and dated informed consent to participate in the study.
- 2. Men or women aged 18 years of age or older of Chinese origin.
- 3. Subjects seeking augmentation therapy for chin retrusion.
- 4. GCRS score of 1 or 2 as assessed by the Blinded Evaluator

#### **Exclusion criteria:**

The presence of any of the following exclusion criteria will exclude a subject from enrolment in the study:

Known/previous allergy or hypersensitivity to any injectable HA gel.

Doc id

Print date:

MA-34970

2023-04-18 09:24

Effective date: 2018-01-15 10:39

- 2. Known/previous allergy or hypersensitivity to local anaesthetics, e.g. lidocaine or other amide-type anaesthetics.
- 3. History of severe or multiple allergies, manifested by anaphylaxis.
- 4. Previous facial surgery, or tissue revitalization treatment with laser or light, needling, mesotherapy, radiofrequency, ultrasound, cryotherapy, chemical peeling or dermabrasion below the level of the horizontal line from subnasale within 6 months before treatment.
- 5. Previous surgery (including aesthetic facial surgical therapy or liposuction), piercing or tattoo in the area to be treated.
- Previous tissue augmentation therapy or contouring with any permanent (non-biodegradable) or semi-permanent filler, autologous fat, lifting threads or permanent implant below the level of the horizontal line from subnasale.
- 7. Previous use of any hyaluronic acid based or collagen based biodegradable facial tissue augmentation therapy in the chin and lips within 12 months before treatment.
- 8. Previous use of any neurotoxin below the level of the horizontal line from subnasale within 12 months before treatment.
- 9. Presence of any disease or lesions near or at the area to be treated, e.g.
  - Inflammation, active or chronic infection (e.g., in mouth, dentals, head and neck region);
  - Facial psoriasis, eczema, acne, rosacea, perioral dermatitis, herpes zoster;
  - Scars or deformities;
  - Cancer or precancer (e.g. actinic keratosis).
- 10. History of radiation or cancer/precancer near or in the area to be treated.
- 11. Subjects with temporomandibular joint dysfunction.
- 12. Subjects with a dental or oral status on visual inspection that in the opinion of the Investigator would make the subject unsuitable for inclusion, or Subjects with dental, oral or sinus surgery within past 6 months prior to the treatment visit or planned such surgery, including dental implants, during the study period.
- 13. History of or active collagen diseases such as systemic lupus erythematosus, rheumatoid arthritis, polymyositis, dermatomyositis, skin or systemic scleroderma.
- 14. Subjects presenting with porphyria.
- 15. Tendency to form keloids, hypertrophic scars, or any other healing disorder.
- History of bleeding disorders or treatment with thrombolytics, anticoagulants or inhibitors of platelet aggregation (e.g. aspirin or other non-steroid anti-inflammatory drugs (NSAIDs), Omega-3, or vitamin E

Effective

Version: 3.0

Effective date: 2018-01-15 10:39

43CH1627 Clinical Study Protocol

Doc id

Print date:

MA-34970

2023-04-18 09:24

GALDERMA

within 2 weeks before treatment.

- 17. Treatment with chemotherapy, immunosuppressive agents, immunomodulatory therapy (e.g. monoclonal antibodies), systemic corticosteroids within 3 months before treatment (inhaled corticoids are allowed).
- 18. Treatment with topical retinoids or corticosteroids on the face below the level of the horizontal line from subnasale within 1 month, or systemic retinoids within 6 months before treatment.
- 19. Any medical condition that in the opinion of the Investigator would make the subject unsuitable for inclusion.
- 20. Other condition preventing the subject from entering the study in the Investigator's opinion, e.g. subjects not likely to avoid other facial cosmetic treatments, subjects anticipated to be unreliable, unavailable or incapable of understanding the study assessments or having unrealistic expectations of the treatment result.
- 21. Women who are pregnant or breast feeding, or Woman of childbearing potential who are not practicing adequate contraception or planning to become pregnant during the study period.
- 22. Subjects planning to accept any other facial plastic surgical or cosmetic procedures below the level of the horizontal line from subnasale during the study (e.g., laser or chemical resurfacing, needling, facelift, radiofrequency etc.).
- 23. Study site personnel, close relatives of the study site personnel (e.g. parents, children, siblings, or spouse), employees, or close relatives of employees at the Sponsor Company.
- 24. Participation in any other clinical study within 30 days before treatment.

## Investigational product,

#### dose and mode of administration:

Restylane Defyne (with lidocaine) consists of stabilized hyaluronic acid of nonanimal origin at a concentration of 20 mg/mL in phosphate buffered saline with lidocaine hydrochloride 3 mg/mL. The study product is supplied in 1 mL syringes. The contents of the syringe are sterile. Two  $27G \times \frac{1}{2}$ " ultra-thin wall needles are co-packed with the syringe for injection.

Restylane Defyne should be injected in the mid to deep dermis, subcutis or supraperiostic zone depending on the area to be treated and the tissue support.

Restylane Defyne will be administered inferior to the lower lip, including the area between the two lines from oral commissure to pre-jowl sulcus.

The injection technique is at the discretion of the Investigator. Other areas in the chin may also be treated to obtain optimal correction. Optimal correction is defined as the best possible aesthetic result that can be obtained for an individual study subject, as agreed upon by the Treating Investigator and subject.

A maximum dosage of 2 mL for Chin Retrusion, and if other areas in the chin are treated for optimal correction, another maximum dosage of 2mL are recommended, at each treatment session, i.e., initial treatment or touch-up treatment respectively.



| Reference therapy,<br>dose and mode of<br>administration: | Not applicable. |
|---|---|
| Duration of treatment and follow-up: | The total duration for each subject will be approximately 14 months for Treatment Group, 20 months for Control Group. |
| Effectiveness Assessment: | Galderma Chin Retrusion Scale (GCRS): |
| | GCRS is a Four-Point scale that assesses the Chin Retrusion from No Retrusion (0) to Severe Retrusion (3) as described below. The Blinded Evaluator and Treating Investigator will rate the subject's Chin for severity of Retrusion using the GCRS at all applicable study visits. |
| | GCRS |
| | No Retrusion: The most anterior portion of the chin is at or near a vertical line drawn from the vermillion border of the lower lip. |
| | Mild Retrusion: The most anterior portion of the chin is clearly recessed, but less than midway, between vertical lines drawn from the vermillion border of the lower lip and the oral commissure. |
| | 2 Moderate Retrusion: The most anterior portion of the chin is recessed approximately midway between vertical lines drawn from the vermillion border of the lower lip and the oral commissure |
| | 3 Severe Retrusion: The most anterior portion of the chin is clearly posterior to the midway point between vertical lines drawn from the vermillion border of the lower lip and the oral commissure. |
| | CCI |

Title
43CH1627 Clinical Study Protocol Doc id ♣ GALDERMA MA-34970

Print date:

2023-04-18 09:24

| | CCI |
|---|---|
| Safety Assessment: | AE will begin to be collected after ICF signed. Each subject will be questioned about AEs at each clinical visit following the screening visit. The question asked will be "Since your last clinical visit have you had any health problems?" Information on AEs can also be obtained from laboratory test report, signs and symptoms detected during each examination, observations by the study personnel, CCI spontaneous reports from the subjects. |
| Statistical Methods: | Primary analysis |
| | The percentage of responders (a responder will be defined as a subject with at least 1 point improvement from baseline GCRS) will be calculated for Treatment Group at 6 months after last treatment, and for Control Group at 6 months after randomization based on the Blinded Evaluator's assessment. In addition, for each group the two-sided 95% confidence intervals around the estimates of the percentage of responders will also be calculated. Secondary analysis The percentage of responders based on the GCRS will also be derived at all applicable follow-up visits for both the Blinded Evaluator's assessment and the Treating Investigator's assessment respectively. The response rates and their 95% confidence interval will be presented by visit and group. |
| | Safety CCI Adverse event incidences will be summarized by MedDRA system organ class (SOC) and preferred term (PT). |
| | Sample size |
| | CCI |

Doc id

Print date:

MA-34970

2023-04-18 09:24

Effective date: 2018-01-15 10:39



Doc id

Print date:

**MA-34970** 

2023-04-18 09:24

# Effective date: 2018-01-15 10:39

## Abbreviations and definitions of terms

AE Adverse Event

Blinded Evaluator An evaluator responsible for independent evaluation of treatment

result(s). The evaluator must not be involved in the treatment of the

subject.

CFDA China Food and Drug Administration

Co-ordinating An Investigator assigned the responsibility for the coordination of Investigator at different centers participating in a multicenter study

CSP Clinical Study Protocol
CTA Clinical Trial Agreement
CTN Clinical trial number
CV Curriculum vitae

Device deficiency Inadequacy of a medical device with respect to its identity, quality,

durability, reliability, safety or performance (includes malfunctions, use

errors, and inadequate labelling)

DMP Data management plan ECG Electrocardiograph

eCRF Electronic Case Report Form

FAS Full Analysis Set

G Gauge

GCP Good Clinical Practice

GCRS Galderma Chin Retrusion Scale

HA Hyaluronic acid

ICF Informed Consent Form

ICH International Conference on Harmonisation

IEC Independent Ethics Committee

IFU Instructions for Use

Investigational Medical device being assessed for safety or performance in a study.

product "Investigational product" is the same as "study device", "investigational

device", or "investigational medical device".

Institution Any public or private entity or agency or medical or dental facility where

clinical studies are conducted.

Investigator The Principal Investigator or other qualified person, i.e. sub-Investigator,

designated and supervised by the Principal Investigator at a study site to perform critical study-related procedures and/or make important study-

related decisions as specified on the delegation log.

Investigator File Essential documents relating to a clinical study as defined in GCP

guidance document and maintained by the Investigator.

LRS Lemperle Rating Scale

Doc id

Print date:

**MA-34970** 

2023-04-18 09:24

MedDRA

Medical Dictionary for Regulatory Activities

**NSAIDs** 

Non-steroid anti-inflammatory drugs

Ы

**Principal Investigator** 

PΡ

Per protocol

QA

Quality assurance Regulatory authority

RAPT

Preferred term

SAE SAP

Serious adverse event Statistical Analysis Plan Source data verification

SDV S-HCG

Serum human chorionic gonadotropin

SOC

System organ class

Sponsor file

Essential documents relating to a clinical study as defined in applicable

GCP guidance document and maintained by the Sponsor.

Study Site

The department of the hospital that participates in the study.

**U-HCG** 

Urinary human chorionic gonadotropin

VLS

Volume Loss Scale

WHO World Health Organization

Effective date: 2018-01-15 10:39

GALDERMA

Title

43CH1627 Clinical Study Protocol

Doc id

MA-34970

# **Table of Contents**

| STUDY ADMINISTRATIVE STRUCTURE | 2 |
|------------------------------------------------------|----------|
| SPONSOR SIGNATURES | 8 |
| SIGNED AGREEMENT OF THE CLINICAL STUDY PROTOCOL | 9 |
| SYNOPSIS | 10 |
| ABBREVIATIONS AND DEFINITIONS OF TERMS | 17 |
| TABLE OF CONTENTS | 19 |
| 1 ETHICAL CONSIDERATIONS | 22 |
| 2 BACKGROUND INFORMATION | 22 |
| 2.1 Indication and population description | 22 |
| 2.2 Investigational product description | 22 |
| 2.3 Reference product description | 23 |
| 2.4 Previous experience | 23 |
| 2.4.1 Non-Clinical Documentation | 23 |
| 2.4.2 Clinical Documentation | 23 |
| 2.5 Study rationale and Justification for design | 24 |
| 2.6 Risk and benefits | 25 |
| 3 OBJECTIVE AND ENDPOINTS | 26 |
| 3.1 Objective of the study | 26 |
| 3.2 Endpoints of the study | 26 |
| 3.2.1 Primary effectiveness endpoint: | 26 |
| 3.2.2 Secondary effectiveness endpoints: | 26 |
| 3.2.3 Safety endpoints: | 26 |
| 4 DESIGN OF THE STUDY | 26 |
| 4.1 General Outline | 26 |
| 4.2 Number of Subjects | 28 |
| 4.3 Duration of Subject Participation | 28 |
| 4.4 Randomization and blinding | 28 |
| 4.4.1 Randomization | 28 |
| 4.4.2 Blinding 4.4.3 Emergency unblinding | 28<br>28 |
| 4.5 Medical history | 28 |
| 4.6 Concomitant Medication, Treatment, and Procedure | 28 |
| 4.7 Schedule of events | 30 |
| 4.8 Visits | 33 |
| 4.8.1 Visits for Group A and Treatment Group | 33 |
| 4.8.2 Visits for Control Group | 34 |
| 5 SUBJECTS | 36 |
| 5.1 Subject information and informed consent | 36 |
| 5.2 Inclusion Criteria | 37 |
| 5.3 Exclusion Criteria | 37 |
| 5.4 Screening and Subject Numbers | 39 |
| 5.5 Withdrawal of Subjects | 39 |



| i itie | | | |
|---------|----------|-------|----------|
| 3CH1627 | Clinical | Study | Protocol |

Doc id

MA-34970

| 6 | STUDY PRODUCTS | 40 |
|---|---|---|
| 6.1 | Investigational Product | 40 |
| 6.2 | Reference Product | 40 |
| 6.3 | Additional Products and Material | 40 |
| 6.4 | Packaging, Labelling and Storage | 40 |
| 6.5 | Product accountability | 41 |
| 6.6 | Treatment | 41 |
| 6.6.1 | | 41 |
| 6.6.2<br>6.6.3 | | 42<br>43 |
| 6.6.4 | | 43 |
| 6.6.5 | , | 43 |
| 6.6.6 | Treatment compliance | 43 |
| 7 | EFFECTIVENESS ASSESSMENTS | 43 |
| 7.1 | General information | 43 |
| 7.2 | Galderma Chin Retrusion Scale (GCRS) | 44 |
| CCI | | |
| 7.5 | Photography | 45 |
| • | | 45 |
| 8<br>CCI | SAFETY ASSESSMENTS | 45 |
| 8.2 | Laboratory assessment | 46 |
| 8.3 | Laboratory assessment | 46 |
| 8.4 | ECG-screening Adverse Events | 40 |
| 8.4.1 | | 47 |
| 8.4.2 | , , | 47 |
| 8.4.3 | Recording Instructions | 47 |
| 8.4.4 | , 3, | 49 |
| 8.4.5<br>8.4.6 | , , , | 49<br>50 |
| 8.4.7 | , , , | 50<br>51 |
| 8.4.8 | • , | 51 |
| 8.5 | Device Deficiencies | 52 |
| 8.5.1 | | 52 |
| 8.5.2<br>8.5.3 | 3 | 52<br>52 |
| 0.5. | | |
| 9 | DATA HANDLING AND MANAGEMENT | 52 |
| 9.1 | Data management | 52 |
| 9.2 | Electronic case report forms | 53 |
| 9.2.1<br>9.2.2 | , | 53<br>54 |
| 9.2.3 | • • • • | 54<br>54 |
| 9.2.4 | , | 54 |
| 9.3 | Source documents | 54 |
| 9.4 | Record keeping and access to source data | 55 |
| 9.5 | Document and data retention | 55 |
| 10 | STATISTICAL METHODS | 55 |
| 10.1 | General | 55 |
| 10.1 | Analysis Populations | 56 |
| 10.2 | Demographics, baseline assessments, and subject characteristics | 56 |
| 10.3 | Effectiveness Analysis | 56 |
| 10.5 | Safety Analysis | 57 |
| 10.6 | | 57 |

| • | 43CH1627 Clinical Study Protocol | Doc id |
|---|---|---|
| GALDERMA | v | MA-34970 |

| 10.7 | Interim Analysis | 58 |
|-------|-------------------------------------------|----|
| 10.8 | Data monitoring committee | 58 |
| 10.9 | Withdrawals and deviations | 58 |
| 10.10 | 0 Sample Size | 58 |
| 11 | PROTECTION OF PERSONAL DATA | 58 |
| 12 | QUALITY CONTROL AND QUALITY ASSURANCE | 59 |
| 12.1 | Quality control | 59 |
| 12.2 | Quality assurance | 59 |
| 12.3 | Changes to the clinical study protocol | 60 |
| 13 | FINANCING, INDEMNIFICATION, AND INSURANCE | 60 |
| 14 | PUBLICATION POLICY | 60 |
| 15 | SUSPENSION OR PREMATURE TERMINATION | 60 |
| 16 | REFERENCES | 62 |
| 17 | APPENDICES | 63 |

# **List of Tables**

| Table 1. | Schedule of Events for Group A and Treatment Group | 30 |
|----------|----------------------------------------------------|----|
| | Schedule of Events for Control Group | |
| Table 3. | Galderma Chin Retrusion Scale | 44 |
| CCI | | |

# **List of Figures**

| Figure 1. | Flow Chart2 | 1 |
|-----------|-----------------|---|
| Figure 2. | Treatment Area4 | 2 |

# **List of Appendices**

| Appendix 1 | Declaration of Helsinki |
|------------|-----------------------------------------------|
| Appendix 2 | Photo guide for Galderma Chin Retrusion Scale |

Doc id

Print date:

2023-04-18 09:24

Effective date: 2018-01-15 10:39

MA-34970

#### **Ethical Considerations** 1

## 1.1 Statement of ethical compliance

The study shall be conducted in compliance with the Clinical Trial Agreement (CTA), the Clinical Study Protocol (CSP), applicable Good Clinical Practice (GCP), and applicable regional or national regulations. The international standard for clinical study of medical devices for human subjects, ISO14155:2011 shall be followed. The International Conference on Harmonisation (ICH) guideline for GCP (E6) shall be followed as applicable for medical device. The study shall be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki (Appendix 1).

### 1.2 Application to independent ethics committee and/or regulatory authorities

It is the responsibility of the Principal Investigator (PI) to obtain approval of the CSP/CSP amendment(s) from the independent ethics committee (IEC). The study shall not begin until the required favourable opinion from the IEC has been obtained. The PI shall file all correspondence with the IEC in the Investigator file and copies of IEC approvals shall be forwarded to the Sponsor. Any additional requirements imposed by the IEC or regulatory authorities (RA) shall be followed.

The collection, access to, processing, and transfer of protected health information or sensitive personal data shall be carried out in accordance with applicable rules and regulations.

#### 2 **Background Information**

#### Indication and population description

As a medical device, Restylane Defyne is intended to augment the volume of facial tissues. In this study, it is intended for the correction of Chin Retrusion in subjects over the age of 18.

#### **Investigational product description** 2.2

Among the different materials used as raw materials in dermal fillers, sodium hyaluronate, also denoted hyaluronic acid when found in vivo and hereinafter referred to as HA, is the most frequently used <sup>1</sup>. Hyaluronic acid is a naturally occurring polysaccharide found in all vertebrates and in some bacteria <sup>1,2</sup>. The chemical structure is very simple with repeating disaccharide units of glucuronic acid and N-acetylglucosamine. As the chemical structure of HA is identical in all species and tissues, it is non-allergenic.

To minimize the risk for contamination, the HA used in the manufacture of Galderma's HA gels is of non-animal source, biosynthesized from Streptococcus species of bacteria. During manufacturing, cross-links are introduced between the HA chains to obtain a gel network and as a result the duration of the gel in the body is several months, as compared to only a few days for a solution of native HA. The HA gel is insoluble in water and organic solvents; however, the gel is highly hydrophilic and swells in water. Hyaluronic acid based fillers typically exhibit better biocompatibility and fewer adverse reactions than fillers based on



other materials. The gel, when injected, acts by increasing the tissue volume, thereby improving tissue structure and support. The gel is gradually degraded over time and eventually the correction made will subside.

Restylane Defyne is a sterile, biodegradable, transparent gel of non-animal cross-linked HA containing a concentration of 20 mg HA per mL in a physiological buffer system. Lidocaine hydrochloride (3 mg/mL) is added to the formulation to diminish the pain resulting from the injection during the treatment. When the gel is injected and the tissue expands some pain can be experienced and it is therefore desirable to have a local anesthetic effect at the site of injection.

Restylane Defyne has been regulatory cleared under the brand name Emervel Deep lidocaine in more than 50 countries from most continents of the world including the US, Europe, Canada, Latin America, Australia, and Asia. The intended use, in the region of origin (Europe), is facial tissue augmentation for the correction of severe wrinkles or to redefine the shape of the face (cheeks, tear troughs, or lips). The regulatory cleared intended use differs between different countries. Depending on the area to be treated and the tissue support, the product should be injected in the mid to deep dermis, submucosal layer of the lips, subcutis, or supraperiostic zone.

The gel in Restylane Defyne is, produced using the Optimal Balance Technology (OBT).

#### 2.3 Reference product description

Not applicable as no dermal filler intended for Chin retrusion correction is available in China at the time of this protocol.

#### 2.4 **Previous experience**

#### Non-Clinical Documentation

Products manufactured using the OBT process have been tested and meet all biocompatibility requirements specified in the international standard ISO 10993:1 (Biological Evaluation of Medical Devices; i.e., having no toxic or injurious effects on the human body) 3,4; it is neither cytotoxic nor genotoxic, and it does not give rise to acute toxicity, pyrogenicity, skin irritation, or delayed sensitization.

In in vivo animal studies, the OBT products demonstrated good filler longevity, similar or superior to comparator products, and all products were well tolerated with minimal microscopic inflammation scores secondary to limited tissue disturbance.

### **Clinical Documentation**

The safety of and performance of Emervel Deep and Restylane Defyne have been evaluated in two randomized controlled studies focusing on nasolabial folds, in one open label study with full-face treatment with the Emervel range of products and in a large observational study.

Restylane Defyne has been evaluated in a 1-year, randomized, evaluator-blinded, active controlled, multi-center, split-face comparison US study of the two HA fillers Restylane Defyne and Juvéderm Ultra Plus with the objective to compare efficacy and safety <sup>12</sup>. One hundred sixty-two (162) subjects with moderate to severe NLFs were treated with Restylane

Doc id

Print date:

**MA-34970** 

2023-04-18 09:24

Defyne in one NLF and Juvéderm Ultra Plus in the other. Non-inferiority of Restylane Defyne compared with Juvéderm Ultra Plus was demonstrated. Restylane Defyne showed a favorable safety profile in subjects with moderate to severe wrinkles and folds, and was comparable to Juvéderm Ultra Plus.

Another randomized, evaluator-blinded study in Europe comparing Emervel Deep (identical to Restylane Defyne but without lidocaine) with Restylane Perlane in 86 subjects, demonstrated similar safety between the dermal fillers and a superior, albeit of limited clinical relevance, efficacy of Emervel Deep after NLF correction <sup>13, 14</sup>.

The performance and safety of the use of Emervel Deep were evaluated for several other indications in an open-label full-face treatment study <sup>6, 15, 16</sup>. These indications included marionette lines (n=92) and tear troughs (n=15). The performance was demonstrated in terms of wrinkle severity improvement and/or aesthetic improvement. In addition, high patient satisfaction was recorded. The improvement was demonstrated to last for up to 6 months for these indications.

In addition, in a large observational study performed in France <sup>8</sup>, 1822 patients were treated with one or more of the Restylane Emervel Collection of products. As it was a non-interventional study product choice and injection volumes were at the discretion of the 58 participating physicians. Emervel Deep was used for several treatment areas including nasolabial folds, marionette lines, tear trough, lip corners, cheek volume, supramental crease, and vertical lip lines. This study investigated mean volumes injected, injection techniques used and tolerance. Performance was not evaluated.

Another Emervel filler products, Restylane Volyme, was evaluated in an 18-month open study17 in 60 subjects with at least Grade 2 on the 4-point volume loss scale (VLS) for full face and at least 2 indications affected among chin, temporal areas, jawline, cheeks, cheekbones, and NLF. Performance was assessed by VLS, Lemperle rating scale (LRS), investigator GAIS, and 3-dimensional (3D) imaging. At 18 months, at least a 1-grade improvement in VLS was observed for full face (68.3% of subjects), chin (77.8%), temporal areas (73.7%), cheeks (66.6%), cheekbones (58.6%), jawline (43.1%), and NLF (71.4%; LRS). For all indications, more than 60% of the volume gained at 3 weeks was sustained at 18 months based on 3D digital imaging. At 18 months, 95.0% of subjects had improved full-face GAIS and all subjects were satisfied with their aesthetic outcome. One subject (1.6%) had treatment-related adverse events.

Post market surveillance data for Restylane Defyne also support that the AE profile is acceptable.

#### 2.5 Study rationale and Justification for design

Chin profile is an important component of the full facial appearance. In Asian people, chin retrusion is very common and many people would like to correct it because chin retrusion may be considered as unattractive. In clinical practice, surgical techniques, such as osteotomy or insertion of implants are commonly used for chin retrusion correction. More recently, HA injection for Chin augmentation has been reported in Chinese people<sup>18, 19</sup>. However, no HA filler intended for Chin Retrusion correction has been approved in China.

Although no published data for Restylane Defyne in Chin retrusion treatment, satisfied outcome was showed in anectdotal report. Also, pre-clinical testing/previous clinical

Doc id 43CH1627 Clinical Study Protocol GALDERMA MA-34970

Print date:

2023-04-18 09:24

experience as described in Section 2.4, have demonstrated acceptable performance and safety for Restylane Defyne when used for facial tissue augmentation. Therefore, the Sponsor consider it justified to conduct a study to investigate Restylane Defyne for the treatment of Chin Retrusion. The study will be used as clinical documentation for registration of the product in China. No treatment control is chosen as no HA filler intended for Chin Retrusion correction is available in China at the time of this protocol.

#### 2.6 Risk and benefits

By January 2017, Restylane Defyne has been regulatory cleared in 50 countries/regions, including US, EU, Canada, Australia, Hong Kong, Korea, India, etc. It is considered safe and effective for facial tissue augmentation.

As all other injectable medical devices, Restylane Defyne has the potential to cause complications. Most events are related to the injected volume and injection technique, though some could be associated with properties or constitutes of the gel itself. After the injection of Restylane Defyne, some common injection-related reactions might occur. These reactions include bruising, erythema, swelling, pain, tenderness, or itching at the implant site. Typically, resolution is spontaneous within one week after injection into the skin. The intensity and duration of these events are usually considered tolerable by a majority of subjects. The study product will be administered in accordance with the instructions in section 6.6.

The primary potential benefit of the study is a perceived improvement in the treated areas. However, there is a risk that the subject will not gain the full aesthetic correction of Chin Retrusion. There is also a risk for development of palpable lumps or displacement of the injected gel. Inflammation or infection have been reported in a few cases after HA filler treatment. There may be risk of damaging body structures such as nerves or blood vessels connected to the injection site, however these risks are minor. Following facial aesthetic treatments isolated rare cases have been reported regarding ischemic events affecting the eye leading to visual loss, and the brain resulting in cerebral infarction. Detailed information on reported AEs relevant for Restylane Defyne is provided in the IB.

Lidocaine can in rare cases give allergic reactions, and therefore subjects with known allergy or hypersensitivity to local anaesthetics should not be included in the study.

The frequency of post market AE reporting is based on the number of units sold. The reporting frequency of AEs assessed as related to Restylane Defyne are ranging from seldom (approximately 1/1 000 - 1/10 000 events per sold unit) to rare/isolated cases (i.e., <1/100 000 events per sold unit).

The risks related to HA filler injections for facial tissue augmentation have been judged to be low, based on nonclinical data (Section 2.4.1), experience from clinical studies (Section 2.4.2) and post-marketing data. Given the anticipated low level of transient and acceptable AEs in connection with the injection, the risk-benefit assessment of the use of Restylane Defyne for treatment of Chin retrusion appears to offer a clinical benefit at reasonable risk.

Only study investigators qualified by education and experience, and who are skilled in the use of dermal fillers from their clinical practice and involvement in clinical research, will be chosen in order to assure proper device implantation and management of study risk.



#### **Objective and Endpoints** 3

#### 3.1 Objective of the study

• To evaluate the effectiveness and safety of Restylane Defyne versus a no-treatment control in the treatment of Chin Retrusion.

#### **Endpoints of the study** 3.2

#### 3.2.1 Primary effectiveness endpoint:

• Percentage of responders, defined by at least 1 point improvement from baseline on the Galderma Chin Retrusion Scale (GCRS), as measured by the Blinded Evaluator at 6 months (after last treatment in Treatment Group, and after randomization in Control Group).

### 3.2.2 Secondary effectiveness endpoints:

- Percentage of responders, defined by at least 1 point improvement from baseline on the GCRS, as measured by the Blinded Evaluator at 3, 9 and 12 months after last treatment in Treatment Group, and at 3 months after randomization, as well as 3, 6, 9 and 12 months after the last treatment in Control Group.
- Percentage of responders, defined by at least 1 point improvement from baseline on the GCRS, as measured by the Treating Investigator at each follow up visit.



## 3.2.3 Safety endpoints:

 Incidence, intensity, duration, and onset of adverse events (AEs) collected throughout the study.



## **Design of the Study**

#### **General Outline** 4.1

This is a randomized, evaluator-blinded, no-treatment controlled study in subjects with Chin Retrusion.

Subjects will be screened for eligibility within 21 days prior to Baseline. Eligible subjects will be randomized either to the Treatment Group or the Control Group in a 3:1 ratio.

Title
43CH1627 Clinical Study Protocol

Doc id

Print date:

MA-34970

2023-04-18 09:24

**Treatment** 

Each subject assigned to the Treatment Group will receive an initial treatment on Day 1. A touch-up treatment may be performed 4 weeks after the initial treatment if optimal chin augmentation has not been obtained. Optimal chin augmentation is defined as the best possible aesthetic result that can be obtained for an individual study participant, as agreed upon by the Treating Investigator and subject. At least one ( $\geq 1$ ) grade improvement from baseline on the GCRS should be the treatment target.

Subjects assigned to the Control Group will not receive treatment at baseline but will return for routine follow-up. At month 6 visit after randomization, subjects in Control Group will be offered a treatment and, at the following visit, an optional touch-up treatment.

## **Evaluation of effectiveness**

Chin Retrusion will be assessed using a separate Four-Point GCRS with photo guides by the Treating Investigator at each visit; and by the Blinded Evaluator at screening, baseline, 3, 6, 9 and 12 months after last treatment in Treatment Group, and at screening, baseline, 3 and 6 months after randomization, as well as 3, 6, 9 and 12 months after last treatment in Control Group.



## **Evaluation of safety**

Information regarding AEs will be collected continuously during the study. CCI



Effective date: 2018-01-15 10:39



#### 4.2 **Number of Subjects**

The study will be performed at approximately 5 sites in China and approximately 148 subjects will be enrolled.

#### **Duration of Subject Participation**

The total duration for each subject will be approximately 14 months for Treatment Group, 20 months for Control Group.

#### Randomization and blinding 4.4

### 4.4.1 Randomization

Approximately 148 subjects will be randomized in a 3:1 ratio to treatment with Restylane Defyne or to no treatment. Before starting the study, a computer generated randomization list will be prepared under the supervision of a designated statistician. The randomization list will be stratified by center.

Each subject will be assigned a subject number as they arrive for the treatment visit. Randomization will be assigned via the eCRF system. The treatment information will be kept by the Treating Investigator during the study not to be disclosed to the Blinded Evaluator.

#### 4.4.2 Blinding

Only the evaluator will be blinded to treatment.

The Blinded Evaluator shall not be allowed to retrieve study supplies or to be present during opening of the study supplies or injections. The Treating Investigator or the subjects are not allowed to discuss treatments with the Blinded Evaluator. All documents with information on study products and randomization assignment shall be kept in a separate binder not available to the Blinded Evaluator.

#### 4.4.3 Emergency unblinding

Not applicable as the Treating Investigator is unblinded.

#### 4.5 **Medical history**

History of surgical events and medical conditions that are judged as relevant by the Investigator shall be documented in the eCRF using medical terminology.

Any concomitant medications and any relevant medical history (including prior facial dermatological procedures performed, and fillers or implants used) or concurrent diseases will be asked for.

#### 4.6 **Concomitant Medication, Treatment, and Procedure**

Except as noted below, concomitant medications or other treatments or procedures may be utilized when the PI or his/her authorized designee considers it medically necessary.

Doc id 43CH1627 Clinical Study Protocol GALDERMA MA-34970

Print date:

2023-04-18 09:24

Information regarding any use of concomitant medications, including over-the-counter medications administered during the study is to be recorded in the eCRF. The generic name or the trade name of all concomitant medication or a description of the procedure and the reason for its use shall be documented in the eCRF.

The following medications, treatments, and procedures are restricted or prohibited during the study:

- Thrombolytics, anticoagulants or inhibitors of platelet aggregation (e.g. aspirin or other non-steroidal anti-inflammatory drugs [NSAIDs]), Omega-3, or Vitamin E should not be used within two weeks before treatment to avoid increased bruising or bleeding at injection sites.
- Lidocaine should be used with caution in patients receiving other local anesthetics or agents structurally related to amide-type local anesthetics e.g., antiarrhythmics, since the systemic toxic effects can be additive.
- Concomitant treatment with chemotherapy, immunosuppressive immunomodulatory therapy (e.g., monoclonal antibodies) is prohibited.
- Long term concomitant treatment with systemic or topical (facial) corticosteroids is prohibited (inhaled corticoids are allowed). Corticosteroids should be used with caution and should be adjudged as necessary by the Investigator.
- Use of systemic or topical (facial) retinoic acid is prohibited.
- Facial tissue augmenting therapy, contouring or revitalization treatment with fillers, lifting threads, permanent implant, needling, mesotherapy, radiofrequency, ultrasound, cryotherapy, fat-injection, neurotoxin, laser or light treatment, chemical peeling or dermabrasion below the level of the horizontal line from subnasale are prohibited.
- Planned surgery including aesthetic facial surgical therapy or facial liposuction, sinus surgery, dental root surgery or dental work, piercing or tattoo in the area to be treated is prohibited.
- Participation in any other clinical study is prohibited

If a subject has used any of the above prohibited medications or performed any of the above prohibited procedures, a protocol deviation will be documented. The subject should continue in the study for the scheduled follow-up visits.



## 4.7 Schedule of events

**Table 2. Schedule of Events for Treatment Group** 

| Treatment Group | | | | | | |
|---|---|---|---|---|---|---|
| | Screening <sup>a</sup> | Baseline <sup>a</sup> /<br>Initial<br>treatment | Optional<br>Touch-up <sup>b</sup> | Follow-up | Follow-up | Final visit / Early termination |
| | D-21 to D1 | D1 | 4W(±3d) after randomization | 4W(±3d) after<br>Last treatment | 3M(±1w), 6M(±1w) and<br>9M (±2w) after last<br>treatment | 12M (±2w) after last<br>treatment |
| Informed consent | X | | | | | |
| Demography | Х | | | | | |
| Medical history & concurrent diseases | х | Х | | | | |
| Concomitant<br>medication/procedures | Х | Х | X | Х | Х | X |
| Vital signs | | Xc | | | | |
| Laboratory tests | Х | | | | Xe | X <sup>f</sup> |
| ECG | Х | | | | | |
| Pregnancy test | X <sup>h</sup> | X <sup>c,i,j</sup> | X <sup>d,i</sup> | | | Xi |
| Inclusion and Exclusion criteria | Х | Х | | | | |
| Randomization | | Х | | | | |
| Treatment | | Х | Х | | | |
| GCRS (Blinded Evaluator) | Х | X <sub>q</sub> | | | Х | Х |
| GCRS(Treating Investigator) | Х | Xq | Xd | Х | Х | Х |
| Photography | | X <sup>d</sup> | Xd | Х | X | Х |

Version: 3.0 Effective Effective Effective

| CCI | | | | | | |
|---------------------|---|---|---|---|---|---|
| Device deficiencies | | Х | Х | | | |
| Assessment of AE | Х | Х | Х | Х | Х | Х |
| Study termination | | | | | | Х |

- a) Screening visit and baseline visit can be combined to one visit if feasible.
- b) This visit is only for subjects who receive touch-up (If no touch-up performed, subjects will conduct the 4w after last treatment visit.
- c) Prior to randomization.
- d) Prior to treatment.
- e) Only performed at 6M.
- f) Only performed at early termination if termination occurs before 6 months visit after last treatment.
- g) Only performed at CC 6M.
- h) Serum pregnancy test (S-HCG).
- i) Urine pregnancy test (U-HCG).
- j) Only performed if the screening S-HCG was done ≥2 weeks before baseline.

**Table 2. Schedule of Events for Control Group** 

| Control Group | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Activity | Screening<br>a | Baseline<br><sup>a</sup> | Follow-up | Follow-up | Follow-up<br>/Treatment | Optional<br>Touch-up <sup>b</sup> | Follow-up | Follow-up | Final visit<br>/ Early<br>termination |
| | D-21 to 1 | D1 | 4W(±3d) after randomization | 3M (±1w) after randomization | 6M(±1w) after randomization | 4W(±3d)<br>after 6M<br>treatment | 4W(±3d)<br>after last<br>treatment | 3M (±1w), 6M(±1w)<br>and 9M (±2w)<br>after last treatment | 12M (±2w)<br>after last<br>treatment |
| Informed consent | Х | | | | | | | | |
| Demography | Х | | | | | | | | |
| Medical history & concurrent diseases | Х | Х | | | | | | | |
| Concomitant medication/procedures | Х | Х | х | х | х | Х | Х | х | Х |
| Vital signs | | Xc | | | Xq | | | | |
| Laboratory tests | Х | | | | Xq | | | Xe | X <sup>f</sup> |

Version: 3.0 Effective Effective Effective

| ♣ GALDERMA | 43CH1627 Clinical Study Protocol | Doe id MA-34970 |
|------------|----------------------------------|-----------------|
|------------|----------------------------------|-----------------|

| Χ | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Xg | X <sup>c,h,i</sup> | | | X <sup>d,h</sup> | X <sup>d,h</sup> | | | X <sup>h</sup> |
| Х | Х | | | | | | | |
| | Х | | | | | | | |
| | | | | Х | Х | | | |
| Х | Х | | Х | Xd | | | Х | Х |
| Х | Х | х | х | Xq | Xq | Х | х | х |
| | Х | Х | Х | Xq | Xd | Х | Х | Х |
| | X X <sup>g</sup> X | X X X X X X X | X X X X X X | X X X X X X X X | X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X <td>X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X</td> <td>X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X</td> | X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X |

| | | | | 1 | 1 | | | 1 | |
|---------------------|---|---|---|---|---|---|---|---|---|
| Device deficiencies | | | | | X | X | | | |
| Assessment of AE | Х | Х | Х | Х | Х | X | Х | X | х |
| Study termination | | | | | | | | | Х |

- a) Screening visit and baseline visit can be combined to one visit if feasible.
- This visit is only for subjects who receive touch-up (If no touch-up performed, subjects will conduct the 4w after last treatment visit).
- Prior to randomization.
- Prior to treatment.
- Only performed at 6M after last treatment
- Only performed at early termination if termination occurs before 6 months visit after last treatment.
- Serum pregnancy test (S-HCG).
- Urine pregnancy test (U-HCG).
- Only performed if the screening S-HCG was done ≥2 weeks before baseline.
- Only performed at CCI 6M after last treatment.

**Effective** 32(63)

Version: 3.0 Effective date: 2018-01-15 10:39

Doc id 43CH1627 Clinical Study Protocol GALDERMA MA-34970

#### 4.8 **Visits**

## 4.8.1 Visits for Treatment Group

### 4.8.1.1 Screening (D-21 to D1)

- Informed consent
- Demography (Initials, Date of birth, Gender and Ethnic origin)
- Screening laboratory tests (haematology and serum chemistry)
- S-HCG for childbearing potential women
- Inclusion and exclusion criteria
- GCRS (by Blinded Evaluator and Treating Investigator)
- Medical history/concurrent diseases including prior facial dermatological procedures performed, and fillers or implants used
- Concomitant medications/procedures
- AE during the visit

#### 4.8.1.2 Baseline (D1)

- Medical history/concurrent diseases
- Vital signs (pulse rate, blood pressure, respiratory rate, body temperature)
- Inclusion and exclusion criteria
- U-HCG for childbearing potential women (Only performed if the screening S-HCG was done ≥2 weeks before baseline)
- Photography (before injection)
- Randomization
- GCRS (by Blinded Evaluator and Treating Investigator)
- Treatment

- Concomitant medications /procedures
- Device deficiencies
- AE since last visit
- 4.8.1.3 Optional Touch-up 4W (±3d) after randomization (only for subjects who receive touch-up)
  - Photography (before injection)
  - GCRS (by Treating Investigator)

- U-HCG for childbearing potential women (before injection)
- Treatment

- Concomitant medications/procedures
- Device deficiencies
- AE since last visit

GALDERMA

Title
43CH1627 Clinical Study Protocol

MA-34970

#### 4.8.1.4 4W ( $\pm 3d$ ) after last treatment

- Photography
- GCRS (by Treating Investigator)



- Concomitant medications /procedures
- AE since last visit

## 4.8.1.5 3M ( $\pm$ 1w), 6M ( $\pm$ 1w) and 9M ( $\pm$ 2w) Follow-up after last treatment

- Photography
- GCRS (by Blinded Evaluator and Treating Investigator)



- Concomitant medications /procedures
- AE since last visit
- Laboratory tests (Only performed at 6M)

#### 4.8.1.6 12M (±2w) after last treatment Final visit or Early termination

- Photography
- GCRS (by Blinded Evaluator and Treating Investigator)

#### CCI

- U-HCG for childbearing potential women
- Concomitant medications/procedures
- AE since last visit
- Laboratory tests (Only performed at early termination if termination occurs before 6 months visit after last treatment)
- Study termination

## 4.8.2 Visits for Control Group

### 4.8.2.1 Screening (D-21 to D1)

- Informed consent
- Demography (Initials, Date of birth, Gender and Ethnic origin)
- Screening laboratory tests (haematology and serum chemistry)
- S-HCG for childbearing potential women
- ECG
- Inclusion and exclusion criteria
- GCRS (by Blinded Evaluator and Treating Investigator)
- Medical history/concurrent diseases including prior facial dermatological procedures performed, and fillers or implants used
- Concomitant medications/procedures
- AE during the visit

#### 4.8.2.2 Baseline (D1)

- Medical history/concurrent diseases
- Vital signs (pulse rate, blood pressure, respiratory rate, body temperature)
- Inclusion and exclusion criteria

GALDERMA

Title
43CH1627 Clinical Study Protocol

MA-34970

- U-HCG for childbearing potential women (Only performed if the screening S-HCG was done ≥2 weeks before baseline)
- Photography
- Randomization
- GCRS (by Blinded Evaluator and Treating Investigator)
- Concomitant medications / procedures
- AE since last visit
- 4.8.2.3 4W (±3d) Follow-up after randomization
  - Photography
  - GCRS (by Treating Investigator)

#### CCI

- Concomitant medications /procedures
- AE since last visit
- 4.8.2.4 3M (±1w) Follow-up after randomization
  - Photography
  - GCRS (by Blinded Evaluator and Treating Investigator)

## CCI

- Concomitant medications /procedures
- AE since last visit
- 4.8.2.5 6M (±1w) Follow-up after randomization / treatment
  - Vital signs (pulse rate, blood pressure, respiratory rate, body temperature)
  - laboratory tests (haematology and serum chemistry)
  - U-HCG for childbearing potential women (before injection)
  - GCRS (by Blinded Evaluator and Treating Investigator)
  - Photography (before injection)

## CCI

Treatment

#### CCI

- Concomitant medications / procedures
- Device deficiencies
- AE since last visit
- 4.8.2.6 Optional Touch-up 4W (±3d) after 6M treatment (only for subjects who received touch-up)
  - Photography (before injection)
  - GCRS (by Treating Investigator)

#### $\mathbb{CC}$

- U-HCG for childbearing potential women (before injection)
- Treatment



GALDERMA

Title

43CH1627 Clinical Study Protocol

MA-34970

- Concomitant medications /procedures
- Device deficiencies
- AE since last visit
- 4.8.2.7 4W (±3d) Follow-up after last treatment
  - Photography
  - GCRS (by Treating Investigator)



- Concomitant medications /procedures
- AE since last visit
- 4.8.2.8 3M ( $\pm 1$ w), 6M ( $\pm 1$ w) and 9M ( $\pm 2$ w) Follow-up after last treatment
  - Photography
  - GCRS (by Blinded Evaluator and Treating Investigator)



- Concomitant medications /procedures
- Laboratory tests (Only performed at 6M)
- AE since last visit
- 4.8.2.9 12M (±2w) after last treatment Final visit / early termination
  - Photography
  - GCRS (by Blinded Evaluator and Treating Investigator)

#### CC

- U-HCG for childbearing potential women
- laboratory tests (haematology and serum chemistry) (Only performed at early termination if termination occurs before 6 months visit after last treatment)
- Concomitant medications /procedures
- AE since last visit
- Study termination

## 5 Subjects

#### 5.1 Subject information and informed consent

The PI or his/her authorised designee must always use the IEC-approved subject information and Informed Consent Form and it must not be changed without prior discussion with the Sponsor and approval from the applicable IEC.

It is the responsibility of the PI or his/her authorised designee to give each subject prior to inclusion in the study, full and adequate verbal and written information regarding all aspects of the clinical study that are relevant to the subject's decision to participate throughout the study, e.g. explain the purpose and procedures of the study, the duration and number of expected participants, possible risks involved, and the opinion of the IEC. The subject shall be informed that the participation is confidential and voluntary and that the subject has the right to withdraw from the study at any time, without any effect on his/her future medical
43CH1627 Clinical Study Protocol

Doc id

Print date:

MA-34970

2023-04-18 09:24

care, treatment or benefits to which the subject is otherwise entitled. The information shall be provided in a language clearly and fully understandable to the subject. The subject shall be given sufficient time to read and understand the Informed Consent Form and to consider participation in the study. Before any study-related activities are performed, the Informed Consent Form shall be personally signed and dated by the subject and the PI or his/her authorised designee responsible for conducting the informed consent process. The consent includes information that data will be collected, recorded, processed, and transferred to countries outside China. The data will not contain any information that can be used to identify any subject.

All signed Informed Consent Forms shall be filed in the Investigator file. The subject shall be provided with a copy of the signed and dated Informed Consent Form and any other written information.

The Investigator shall ensure that important new information is provided to new and existing subjects throughout the study

#### 5.2 Inclusion Criteria

The subject must meet the following criteria to be eligible for the study:

- 1. Signed and dated informed consent to participate in the study.
- 2. Men or women aged 18 years of age or older of Chinese origin.
- 3. Subjects seeking augmentation therapy for chin retrusion.
- 4. GCRS score of 1 or 2 as assessed by the Blinded Evaluator.

#### 5.3 Exclusion Criteria

The presence of any of the following exclusion criteria will exclude a subject from enrolment in the study:

- 1. Known/previous allergy or hypersensitivity to any injectable HA gel.
- 2. Known/previous allergy or hypersensitivity to local anaesthetics, e.g. lidocaine or other amide-type anaesthetics.
- 3. History of severe or multiple allergies, manifested by anaphylaxis.
- 4. Previous facial surgery, or tissue revitalization treatment with laser or light, needling, mesotherapy, radiofrequency, ultrasound, cryotherapy, chemical peeling or dermabrasion below the level of the horizontal line from subnasale within 6 months before treatment.
- 5. Previous surgery (including aesthetic facial surgical therapy or liposuction), piercing or tattoo in the area to be treated.
- 6. Previous tissue augmentation therapy or contouring with any permanent (non-biodegradable) or semi-permanent filler, autologous fat, lifting threads or permanent implant below the level of the horizontal line from subnasale.

Effective date: 2018-01-15 10:39

43CH1627 Clinical Study Protocol

Doc id

Print date:

**MA-34970** 

2023-04-18 09:24

7. Previous use of any hyaluronic acid based or collagen based biodegradable facial tissue augmentation therapy in the chin and lips within 12 months before treatment.

- 8. Previous use of any neurotoxin below the level of the horizontal line from subnasale within 12 months before treatment.
- 9. Presence of any disease or lesions near or at the area to be treated, e.g.
  - Inflammation, active or chronic infection (e.g., in mouth, dentals, head and neck region);
  - Facial psoriasis, eczema, acne, rosacea, perioral dermatitis, herpes zoster;
  - Scars or deformities;
  - Cancer or precancer (e.g. actinic keratosis).
- 10. History of radiation or cancer/precancer near or in the area to be treated.
- 11. Subjects with temporomandibular joint dysfunction.
- 12. Subjects with a dental or oral status on visual inspection that in the opinion of the Investigator would make the subject unsuitable for inclusion, or Subjects with dental, oral or sinus surgery within past 12 months prior to the treatment visit or planned surgery, including dental implants, during the study period.
- 13. History of or active collagen diseases such as systemic lupus erythematosus, rheumatoid arthritis, polymyositis, dermatomyositis, skin or systemic scleroderma.
- 14. Subjects presenting with porphyria.
- 15. Tendency to form keloids, hypertrophic scars, or any other healing disorder.
- 16. History of bleeding disorders or treatment with thrombolytics, anticoagulants or inhibitors of platelet aggregation (e.g. aspirin or other non-steroid anti-inflammatory drugs (NSAIDs), Omega-3, or vitamin E within 2 weeks before treatment.
- 17. Treatment with chemotherapy, immunosuppressive agents, immunomodulatory therapy (e.g. monoclonal antibodies), systemic corticosteroids within 3 months before treatment (inhaled corticoids are allowed).
- 18. Treatment with topical (facial below the level of the horizontal line from subnasale) retinoids or corticosteroids within 1 month, or systemic retinoids within 6 months before treatment.
- 19. Any medical condition that in the opinion of the Investigator would make the subject unsuitable for inclusion.
- 20. Other condition preventing the subject from entering the study in the Investigator's opinion, e.g. subjects not likely to avoid other facial cosmetic treatments, subjects anticipated to be unreliable, unavailable or incapable of understanding the study assessments or having unrealistic expectations of the treatment result.

Effective date: 2018-01-15 10:39

- 21. Women who are pregnant or breast feeding, or Woman of childbearing potential who are not practicing adequate contraception or planning to become pregnant during the study period.
- 22. Subjects planning to accept any other facial plastic surgical or cosmetic procedures below the level of the horizontal line from subnasale during the study (e.g., laser or chemical resurfacing, needling, facelift, radiofrequency etc.).
- 23. Study site personnel, close relatives of the study site personnel (e.g. parents, children, siblings, or spouse), employees, or close relatives of employees at the Sponsor Company.
- 24. Participation in any other clinical study within 30 days before treatment.

### 5.4 Screening and Subject Numbers

Each screened subject will be assigned a screening number consisting of "S" and the site number followed by a consecutive number starting with 01 at each site, e.g. S101, S102. The screening number shall be listed on a subject screening and inclusion log.

A "screening failure" is defined as a subject who does not fulfil the eligibility criteria. For screening failures, the eCRF screening visit shall be completed to an extent that makes it clear which assessments have been made and the reason why the subject did not fulfil the eligibility criteria. The reason for excluding a subject from entering the study shall also be specified in the subject screening and inclusion log.

When the Investigator has confirmed that all inclusion criteria and no exclusion criteria are met, each enrolled subject will be assigned a subject number by the eCRF, consisting of the site number followed by a consecutive number starting with 001 at each site, e.g. 1001, 1002.

The subject number, subject name, and other information sufficient to link the eCRF to the medical records (e.g. national identification number, chart number, etc.) shall be recorded on a subject identification list. The subject identification list shall only be available at the site, both throughout and after the study.

#### 5.5 Withdrawal of Subjects

Each subject shall be advised in the Informed Consent Form that the subject has the right to withdraw from the study at any time, for any reason, without prejudice. Subjects may also be discontinued from this study if the Investigator determines that it is in the subject's best interest to do so, and may be withdrawn at the Investigator's discretion at any time. The withdrawal criteria are:

- Medical reasons: If the subject suffers from a medical condition that in the judgement
  of the Investigator makes it medically necessary to withdraw the subject. The specific
  rationale for Investigator-initiated withdrawal of a subject for medical reasons shall
  document the specific condition for withdrawing the subject.
- **Withdrawal of informed consent:** A subject can withdraw their consent to participate in the study at their own request or be withdrawn from participation in the study at the request of their legally authorised representative at any time for any reason.

Doc id 43CH1627 Clinical Study Protocol GALDERMA MA-34970

- Lost to follow-up: If a subject does not return for a scheduled visit, reasonable effort shall be made to contact that subject, e.g. call three times at different hours and leave messages if applicable before declaring the subject lost to follow-up.
- Other: Examples of other reasons for withdrawal may be failure to comply with protocol requirements or to complete the protocol-specified evaluations.

The reason and date for withdrawal shall be documented in the eCRF. When possible, an explanatory comment shall be added in the study termination module/pages to further explain the reason for withdrawal. If withdrawal of a subject occurs during a regular study visit, the eCRF for that specific visit shall be completed as far as possible together with the study termination eCRF module.

If withdrawal of a subject occurs between regular study visits the subject should when possible (irrespective of the reason for withdrawal) be scheduled for a termination visit. In these cases the eCRF for the early termination visit should be completed. The subject will need to follow the same requirements for the final visit.

If a subject is withdrawn from the study, all data collected until the time of withdrawal will be used in the analyses.

A withdrawn or discontinued subject must not be replaced or re-entered into the study.

If an AE which, according to the Investigator's assessment, is related to the use of any of the study products and is still ongoing at the time of the withdrawal, such events shall be followed-up after the last study visit until resolved, assessed as chronic or stable, or for at least three months.

#### 6 Study Products

#### 6.1 **Investigational Product**

Restylane Defyne (with lidocaine) consists of stabilized hyaluronic acid of non-animal origin at a concentration of 20 mg/mL in phosphate buffered saline with lidocaine hydrochloride 3 mg/mL. The study product is supplied in 1 mL syringes. The contents of the syringe are sterile. Two 27G × ½" ultra-thin wall needles are co-packed with the syringe for injection.

#### 6.2 **Reference Product**

Not applicable.

#### **Additional Products and Material** 6.3

The study product is supplied in 1 mL syringes with sterile contents, together with two 27G × ½" Ultra thin wall needles for injection. Any other materials will be supplied by the site.

#### Packaging, Labelling and Storage 6.4

Restylane Defyne is manufactured by Q-Med AB, Uppsala, Sweden who will supply the study products. Restylane Defyne, commercially available in EU, will be used for the study.

The syringes are labelled with name of the product, name of the manufacturer (Q-Med AB). The syringe and needles are packed in a blister and put in a carton. The carton will be

labelled in local language, specifying the protocol number, lot number, expiry date and that the product is to be used for clinical studies exclusively.

The study products should be stored at a temperature up to 25°C and protected from sunlight and freezing. Opened syringes should not be re-used. Accountability will be performed as specified in section 6.5.

#### 6.5 Product accountability

The study product will be released to the PI or his/her authorised designee after study approvals have been received from the IEC and the CTA has been signed by all parties.

The PI must ensure that the study product is kept in a secure location, with access limited to those authorised by the PI.

The study product must be traceable from the manufacturer to its use in subjects until return or disposal. It is therefore important that the PI maintains accurate product accountability records, i.e. documentation of the physical location of all study product, deliveries, and return of study product between the Sponsor or a third-party vendor and the PI, and documentation of administration of product to the subject. A shipping record shall be kept of all study products received from the Sponsor; including the product name, date received, batch number, expiration date, and amount received. In addition, dispensing logs shall be maintained including the product name, dispense date, the number of syringes used, the number of syringes left in stock, and the subject receiving study product. A log for accountability procedure is provided by the Sponsor.

When the study is completed, all unused or expired study product at each study site shall be returned to the Sponsor or a third-party vendor for destruction. Any malfunctioning study products shall be reported as described in Section 8.5.3.

Product deliberately or accidentally destroyed during shipment or at a study site shall be accounted for and documented. Used syringes, disposable needle, and any opened unused material must be discarded and must not be reused according to standard procedures at the site. Disposal of hazardous material, i.e. syringes and needles must conform to applicable laws and regulations. The study product must not be used outside the study.

#### 6.6 Treatment

#### 6.6.1 <u>Treatment Procedure</u>

The subjects will be informed about the indications, expected result, precautions, and potential AEs.

Injection procedures are associated with a risk of infection. Aseptic technique and standard practice to prevent cross-infections should be observed at all times including the use of disposable gloves during the injection procedure. The subject should not wear make-up that might affect the treatment or evaluation on the day of treatment, if such make-up was already applied this must be completely removed prior to any injection. The treatment site should be thoroughly cleaned at least twice with a suitable antiseptic solution.

Restylane Defyne should be injected in the mid to deep dermis, subcutis or suprapriostic zone depending on the area to be treated and the tissue support. .

Doc id



43CH1627 Clinical Study Protocol

MA-34970

Restylane Defyne will be administered inferior to the lower lip, including the area between the two lines from oral commissure to pre-jowl sulcus (Figure 2).

Figure 2. Treatment area



The injection technique is at the discretion of the Investigator. One potential injection technique includes administration of Restylane Defyne at one injection point at the most anterior portion of the chin with or without 2 points (one per side) on the sides of the chin for certain subjects based on the discretion of investigators. Other areas in the chin may also be treated to obtain optimal correction. Optimal correction is defined as the best possible aesthetic result that can be obtained for an individual study subject, as agreed upon by the Treating Investigator and subject.

To avoid breakage of the needle, no attempt to bend or otherwise manipulate the needle before or during treatment is recommended. Before injecting, the air should be removed by pressing the rod carefully until a small droplet is visible at the tip of the needle. Aspiration prior to injection in order to avoid accidental intravascular injection is recommended.

Injection should stop just before the needle is pulled out from the skin to prevent material from leaking out from the injection site. Excessive pressure must not be applied at any time during injection. If resistance is encountered the needle should be partially withdrawn and repositioned or fully withdrawn and checked for function. The injection sites may be gently massaged by the Treating Investigator to conform the contour of the surrounding tissue.

### Treatment regimen (dose)

A maximum dosage of 2 mL for Chin Retrusion, and if other areas in the chin are treated for optimal correction, another maximum dosage of 2mL are recommended, at each treatment session, i.e., initial treatment or touch-up treatment respectively.

#### 6.6.3 Post-treatment Care

Ice in appropriate packaging can be applied on the treatment site for a short period to reduce swelling and discomfort.

After the injection, some common injection-related reactions might occur. These reactions include erythema, swelling, pain, itching, bruising or tenderness at the implant site. Typically, resolution is spontaneous within one week after injection into the skin. The patient must avoid exposing the treated area to heat (sun bathing, sauna, steam baths, etc.) or extreme cold least until any initial swelling and erythema has resolved. In order to prevent infections, the patient should avoid touching the treated area and no creams or cosmetics should be applied before the skin has healed completely.

#### 6.6.4 Post-trial provisions

After the study is finalised Q-Med AB will not supply any more treatments to the subjects, even if the result does not persist.

## 6.6.5 Electronic case report form recordings

The following details of each injection are to be recorded in the eCRF:

- Date for administration
- Lot number
- Local anaesthetic used (product name, volume injected/amount applied, and concentration)
- Administered volume (for chin retrusion and other areas in the chin for optimal correction)
- Injection technique (retrograde/anterograde line injection, etc)
- Depth of injection
- Post-treatment care (massage, ice pack, etc)

In addition, any technical problems (device deficiencies) or clinical complications (AEs) associated with the injection will be recorded in the eCRF.

### 6.6.6 <u>Treatment compliance</u>

The treatment is an implant administered by the Treating Investigator and the details of the administration are recorded in the eCRF. No other measurements of treatment compliance will be made.

#### 7 Effectiveness Assessments

#### 7.1 General information

The methods for collecting effectiveness data include assessment of GCRS <sup>9</sup>(Section 7.2),

A description of the laboratory assessments is given in Section 8.2 and the ECG assessment in Section 8.3.

Assessments will be performed by CCI , the Treating Investigator, and the Blinded Evaluator, as described in the respective section. To avoid inter-observer variability, every



effort should be made to ensure that preferably the same individual who made the initial baseline determinations completes all corresponding follow-up evaluations. If it is not possible to use the same evaluator/investigator to follow the subject, evaluations should be overlapped (examine the subject together, discuss findings, and both sign in souce data) for at least 1 visit.

#### 7.2 Galderma Chin Retrusion Scale (GCRS)

GCRS is a validated Four-Point scale assesses the Chin Retrusion from no retrusion (0) to severe retrusion (3) as described below. A validation study concluded that the accuracy of this assessment tool was acceptable for use in assessing correction of Chin Retrusion in live assessment of subjects9. The Blinded Evaluator will rate the subject's Chin Retrusion using the GCRS at screening, baseline, 3, 6, 9 and 12 months after last treatment in Treatment Group; and at screening, baseline, 3 and 6 months after randomization, as well as 3, 6, 9 and 12 months after last treatment in Control Group. The Treating Investigator will do the GCRS evaluation at all visits in each group. The Blinded Evaluator and Treating Investigator will conduct their GCRS assessments using a photoguide (Appendix 2). During the GCRS assessment, the subject shall have a neutral facial expression; with the head in an upright position and look straight at eye level with closed and relaxed lips.

Table 3. Galderma Chin Retrusion Scale

| GCRS | |
|---|---|
| 0 | No Retrusion: The most anterior portion of the chin is at or near a |
| | vertical line drawn from the vermillion border of the lower lip. |
| 1 | Mild Retrusion: The most anterior portion of the chin is clearly |
| | recessed, but less than midway, between vertical lines drawn from |
| | the vermillion border of the lower lip and the oral commissure. |
| 2 | Moderate Retrusion: The most anterior portion of the chin is |
| | recessed approximately midway between vertical lines drawn from |
| | the vermillion border of the lower lip and the oral commissure |
| 3 | Severe Retrusion: The most anterior portion of the chin is clearly |
| | posterior to the midway point between vertical lines drawn from the |
| | vermillion border of the lower lip and the oral commissure. |





## 7.5 Photography

Digital photographs will be taken of each subject pre-treatment at visits when treatment is performed and at each follow-up visit. The photographs will be used to document condition during the study; CCI . If necessary, the photo should be taken when AEs occur to document AEs in the treated area. Note that no make-up that might affect the treatment or evaluation should be used on the photographs.

Each Investigator and other study site personnel designated to take photographs, if applicable, shall be thoroughly trained in the equipment and techniques, and how to upload photographs to the secured web portal, if applicable, before study start. The same photographic equipment and standardized setting must be used at each visit (e.g., distance, light, facial position and expression). For further details, please see the instruction of image procedures in the photo user guide.

All photos should be taken from a straight frontal view and both lateral views with full face frame. The subject shall have a neutral facial expression; with the head in an upright position and look straight at eye level with closed and relaxed lips.

Each photograph shall be labelled with the subject initials, subject number, as well as the visit ID and visit date at which the photograph was taken. In order to maintain Confidentiality, the photographs must not include any information that may reveal the subject's identity.

# 8 Safety Assessments





#### 8.2 Laboratory assessment

Laboratory samples will be taken at the screening visit (day -21 to day 1), at 6 months visit after last treatment or at early termination if termination occurs before 6 months visit after last treatment for all subjects. In Control Group, it will also be taken at 6 months visit before treatment.

The following laboratory assessments will be performed:

- Haematology: haemoglobin, red blood cells, white blood cells, differential count and platelet count.
- Serum chemistry: renal function tests (creatinine and BUN); and liver function tests (aspartate amino transferase (ASAT), alanine amino transferase (ALAT) total bilirubin and direct bilirubin).

A serum pregnancy test (S-HCG) in women of childbearing potential will be performed at screening. A urine pregnancy test (U-HCG) in women of childbearing potential will be performed prior to randomization at baseline, if the screening S-HCG was done ≥2 weeks before the baseline visit, prior to 6M treatment (only for Control Group), prior to touch-up treatment, and at the study completion or early termination. The results of the hematology and serum chemistry will only be used for safety assessment by investigator and will not be collected in the eCRF. The pregnancy test results for women of childbearing potential will be recorded in the eCRF.

Other laboratory test might be performed at the discretion of the investigator. All laboratory assays will be performed at a local laboratory. Reference ranges will be supplied by the laboratory and used by the Investigator to assess the laboratory data for clinical significance and out of range pathological changes.

Any clinical significant abnormal laboratory values at the 6 months visit after last treatment or early termination visit will be reported as AEs in the eCRF. In the control group, clinical significant abnormal laboratory values at the 6 months visit after randomization will also be reported as AEs.

#### 8.3 ECG-screening

ECG will be taken at the screening visit (day -21 to day 1) and assessed by investigator for clinical significance. The results of ECG will only be used for screening purposes by the investigator and will not be collected in the eCRF.

Effective date: 2018-01-15 10:39

43CH1627 Clinical Study Protocol

Doc id

Print date:

MA-34970

2023-04-18 09:24

# 8.4 Adverse Events

## 8.4.1 Definition of Adverse Events

An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons\*, whether or not related to the study product.

This definition includes:

- events related to the investigational product or the reference product
- events related to the procedures involved

#### 8.4.2 Definition of Serious Adverse Event

A serious adverse event (SAE) is an AE that:

- a) led to death,
- b) led to serious deterioration in the health of the subject, that either resulted in
  - 1. a life-threatening\*\* illness or injury, or
  - 2. a permanent impairment of a body structure or body function, or
  - 3. in-patient or prolonged hospitalisation\*\*\*, or
  - 4. medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function,
- c) led to foetal distress, foetal death, or a congenital abnormality or birth defect

In cases of doubt, whether an AE fulfils a serious criterion or not, there should be a predisposition to report as a SAE rather than not report as such (see section 8.4.4).

#### 8.4.3 Recording Instructions

AE will begin to be collected after ICF signed. Each subject will be questioned about AEs at each clinical visit following the screening visit. The question asked will be "Since your last clinical visit have you had any health problems?" Information on AEs can also be obtained from signs and symptoms detected during each examination or from a laboratory test, observations by the study personnel, spontaneous reports from the subjects.

When an AE is related to a device deficiency (refer to section 8.5), including technical device malfunction, the AE shall be recorded on the AE module in the eCRF and the technical complaint shall be reported separately on the clinical study complaint form.

Investigators, or other study personnel, will record all AEs in the eCRF, including:

<sup>. \*</sup>For users or other persons, this definition is restricted to events related to the investigational product

<sup>\*\*</sup>The term "life-threatening" in the definition of "serious" refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe. (Source: ICH-E2A clinical safety data management: definitions and standards for expedited reporting).

<sup>\*\*\*</sup> Planned hospitalisation for a pre-existing condition, or a procedure required by the CSP, without serious deterioration in health, is not considered a SAE. (Source: ISO14155:2011).

- Event term (recorded in standard medical terminology and avoiding abbreviations),
- Description of event and affected area (if applicable),
- Start date (First day with symptoms)
- Stop date (Last day with symptoms)
- Intensity (mild, moderate or severe according to definition in section 8.4.3.1)
- Seriousness (serious or not serious, according to definition in section 8.4.2)
- Causal relationship to study product and study product injection procedure (yes or no)
- Action taken (none, medication treatment, non-pharmacological treatment or other procedures/ tests, subject withdrawn)
- Outcome of the AE (ongoing, recovered, recovered with sequelae, death, chronic/ stable, not recovered at study end)

The AE module in the eCRF must be signed and dated by the Investigator.

#### 8.4.3.1 Intensity

For each reported AE, the intensity will be recorded. The following definitions of intensity are to be used:

Mild: A mild AE means awareness of symptoms or signs, but easily tolerated

(acceptable).

**Moderate:** A moderate AE means enough discomfort to interfere with usual activity

(disturbing).

**Severe:** A severe AE means incapacity to work or to do usual activity

(unacceptable).

If the intensity changes over time the maximum intensity of the AE should be recorded.

#### 8.4.3.2 <u>Causal Relationship and Seriousness</u>

Each AE, serious as well as non-serious, will be assessed by the Investigator for causal relationship with the study product and its use (the injection procedure) and for seriousness (yes or no) of the event.

A two-point scale (Yes or No) will be used for causality assessments. The Investigators shall be asked to indicate a response to each of the following questions in the eCRF:

- "Do you consider that there is a reasonable possibility that the event may have been caused by the study product?" and
- "Do you consider that there is a reasonable possibility that the event may have been caused by the study *product injection procedure*?"

If any of these questions is answered Yes, the AE is considered related. There may be events that are only related to product or procedure.



Each AE will also be assessed for causal relationship and seriousness by the Sponsor, in order to fulfil regulatory requirements.

#### **Reporting of Adverse Events**

AE reporting on each subject will start after the ICF has been signed. The reporting will continue during each follow-up visit (including telephone contacts and extra visits between planned visits) until the last scheduled visit in the study.

All AEs, non-serious as well as serious, are to be reported as an AE in the eCRF.

## **Reporting of Serious Adverse Events**

After aware of any SAE, the Investigator shall report it to his/her administrative department of medical device clinical trials under the clinical trial institution, which in turn shall notify the Sponsor Representative in writing. This initial report can be made via fax or e-mail or submitted via the eCRF.

In case of difficulty to obtain all the required information within 24 hours, an initial report can be submitted, with the following information as a minimum, irrespective of whether some of it is regarded as preliminary:

- CTN
- Subject identification (age, gender, subject number)
- AE description
- date when AE occurred
- date when AE became serious
- Name of PI and original reporter (if other than Investigator)
- Name of study product
- Treatment specification

The Investigator will assure completeness of the SAE information and the supporting documentation.

Follow-up information and data missing in the initial SAE reporting shall be gathered as soon as possible and reported to the Sponsor via Sponsor's representative immediately but not later than 24 hours of awareness of the new data. Complete and adequate information on each SAE is required. All attempts to obtain this information, including dates for follow-up activities, must be documented by the Investigator.

### Supporting documentation to be provided with the SAE report:

- Concomitant Medication Form/list
- Concomitant Procedure/Treatment Form/list
- AE Form/list
- Medical History Form/list



 Any other relevant supporting documentation (e.g. hospital notes, death certificate, autopsy reports etc.)

\_\_\_\_\_

Fax number for SAE reporting: +46 18 474 91 01

**E-mail for SAE reporting:** safety.q-med@galderma.com

Surface mail for providing

complementary information: Q-Med AB

Attn. Corporate Medical Affairs & Vigilance

Seminariegatan 21

SE-752 28 UPPSALA, Sweden

E-mail for Device deficiency,

Clinical Study Complaint Form: Complaints.q-med@galderma.com

\_\_\_\_\_

E-mail address will be pre-programmed in the eCRF system.

For non-urgent complementary information not possible to send by e-mail or fax, please use surface mail.

The SAE form (CFDA template in Chinese) must be signed and dated by the Investigator. If the initial 24-hour SAE report does not contain full information or if it is made without using the SAE form, the fully completed and signed SAE form shall be e-mailed or faxed to the Sponsor (contact details refer to 24-hour contact person list in ISF). A copy of the fully completed SAE form shall be kept at the site.

In addition, according to national regulations, the investigator will report a SAE Form (CFDA SAE template) to the administrative department of medical device clinical trials in his/her hospital, and they should, within 24 hours, deliver a written report to the corresponding Ethics Committee and the local food and drug administrative department of province, autonomous region and municipality at the place where the clinical trial institution locates. In case of a death incident, the clinical trial institutions and investigators should furnish the Ethics Committee and the Sponsor Representative with all required materials.

The Sponsor Representative in China is responsible for, within five (5) business days upon being informed, reporting any SAE or device defect with the likelihood of SAE to Shanghai Municipal FDA and Shanghai Municipal Commission of Health and Family Planning by fax or mail. The relevant correspondence will be documented in TMF; meanwhile, the Sponsor Representative should notify other clinical trial institutions and investigators participating in the study, and promptly report it to the Ethics Committee of the involved clinical trial institutions via the administrative department of medical device clinical trials according to national regulations.

# 8.4.6 Follow-up of Unresolved Events after study termination and new Events after study termination.

All serious as well as non-serious AEs with a causal relationship to the study product or treatment procedure and ongoing at study end, shall be followed up after the subject's



Print date:

2023-04-18 09:24

participation in the study is over. Such events shall be followed-up after the last study visit until resolved, assessed as chronic or stable, or for at least three months. Final outcome after study end should be reported on a paper AE form.

All serious as well as non-serious AEs with a causal relationship to the study product or treatment procedure with onset after subject participation in the study has ended that the investigator become aware of, shall be collected and reported to Sponsor on a paper AE form or in the post marketing AE form or SAE paper form if applicable. The events shall thereafter be followed up until resolved or considered chronic or stable, or for at least three months. Final outcomes shall be reported on the AE follow up form or in the post marketing AE form. The Investigator shall report any such AE or SAE including all previous Adverse events reported during the study and medical history of the patient to the Sponsor immediately but not later than 24 hours of awareness of the event. This report can be made via fax or e-mail according to contact details specified in section 8.4.5.

#### 8.4.7 Pregnancy

Pregnancy itself is not regarded as an AE.

If there is a pregnancy during the study period the subject must continue to be followed within the study and the outcome of pregnancy must be reported even if the expected date of delivery occurs after study completion.

A pregnancy confirmed during the study period must be reported by the Investigator on a pregnancy report form immediately upon acknowledge be submitted to the Sponsor according to contact details specified in section 8.4.5. The report can be prospective or retrospective. Follow-up shall be conducted to obtain outcome information on all prospective reports.

Cases that led to foetal distress, foetal death or a congenital abnormality or birth defect are to be regarded as SAEs and shall be reported on the exposure *in utero* report form to the Sponsor immediately but no later than 24 hours after the Investigators awareness. These events shall be handled as SAEs during data processing. Other complications during the pregnancy that are related to the pregnant woman and fulfils any serious criteria, such as pre-eclampsia requiring hospitalisation, shall be reported and handled as SAEs. Elective abortions without complications will not be reported as AEs.

## 8.4.8 Anticipated Adverse Events

After the injection some common injection-related reactions might occur with both products. These reactions include bruising, erythema, swelling, pain, tenderness and itching at the injections site. Typically these reactions start on the day of treatment and resolve spontaneous within one week after injection, as observed in the Chinese clinical study for Restylane and in consistent with international results for both products.

Refer to the Restylane Defyne IB for all anticipated AEs.



#### 8.5 **Device Deficiencies**

#### Definition of Device Deficiency 8.5.1

A device deficiency is defined as an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety\* or performance.

Note: Device deficiencies include malfunctions, use errors, and inadequate labelling.

\*Inadequacy of device safety refers to properties of the device which could have or have led to an AE.

#### **Recording Instructions** 8.5.2

When a device deficiency is discovered the Clinical Study Complaint Form in the eCRF will be completed by the Investigator. The type of complaint shall be described and injury to the subject or user or unintended exposure to study product shall be reported as applicable. If an injury has occurred, an AE module or a SAE Form should be completed following instructions in section 8.4. If no SAE was experienced as a result of the device deficiency the Investigator shall assess whether or not the device deficiency could have led to an SAE if:

- Suitable action had not been taken,
- Intervention had not been made or,
- Circumstances had been less fortunate

The Sponsor will also make the same assessment in the Clinical Study Complaint Form.

#### Reporting Device Deficiency

The Investigator will complete the Clinical Study Complaint Form to the Sponsor using the contact details specified in section 8.4.5. A device deficiency that led to a SAE and any device deficiency that could have led to a SAE shall be reported within 24 hours after the Investigator's awareness in accordance to section 8.4.5.

In order to fulfil regulatory reporting requirements, all deficiencies with the study product must be assessed by both the Investigator and the Sponsor to determine if it could have led to a SAE. This assessment will be documented in the Clinical Study Complaint Form.

If an SAE has resulted from a device deficiency or if either the Investigator or the Sponsor assesses that the device deficiency could have led to an SAE the event will be reported in accordance with Regulatory requirements, as applicable.

The deficient study product shall be kept, if applicable, by the study site until the QA complaints group has confirmed whether the product shall be returned to Sponsor for further study or if it can be destroyed at the study site.

#### 9 **Data Handling and Management**

## **Data management**

Data management based on GCP refers to the activities defined to achieve safe routines to enter clinical data information into a database, efficiently and avoiding errors. The data management routine includes procedures for handling eCRFs, database set-up and 43CH1627 Clinical Study Protocol

Doc id

Print date:

MA-34970

2023-04-18 09:24

Effective date: 2018-01-15 10:39

Effective

management, data entry and verification, data validation, and documentation of the performed activities including information of discrepancies in the process. The data management process will be described in detail in the data management plan (DMP).

The database, the data entry screens and program will be designed in accordance with the CSP. Data validation will be performed by computerised logical checks and manual review. Drugs and events will be coded in accordance with World Health Organization (WHO) Drug and medical dictionary for regulatory activities (MedDRA) dictionaries as specified in the DMP. Safety data (SAE) in the clinical database will be reconciled against the data in the safety database.

When all efforts have been made to ensure that the data recorded in the eCRFs and entered in the database is as correct and complete as possible, the clinical database will be locked. Study data will be transferred to SAS datasets which thereafter will be write-protected. Statistical analyses will be generated in SAS using data from the locked datasets.

## 9.2 Electronic case report forms

An eCRF is required and shall be completed electronically for each screened subject (screening visit) and included subjects (subsequent visits).

The eCRF includes password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate. Study data will be transcribed directly from the source documents, which are to be defined at each site before inclusion of the first subject.

Authorised study site personnel designated by the PI shall complete data collection. Appropriate training and security measures shall be completed with all authorised study site personnel prior to the study being initiated and any data being entered into the system for any subject.

The study data is the sole property of the Sponsor and shall not be made available in any form to third parties without written permission from the Sponsor. At the end of the study, electronic data are kept at the Sponsor and a copy (provided by the vendor) at the study site as part of the Investigator file.

Any delegation of collection of data shall be specified in a signature and delegation log.

#### 9.2.1 Data entry

All data shall be entered in English. The eCRFs should always reflect the latest observations on the subjects participating in the study. Therefore, the eCRFs shall be completed within 5 working days after the subject's visit. The subject's identity must always remain confidential, i.e. the name and address of the subjects must not be registered in the eCRFs or in the database. The Investigator must verify that all data entries in the eCRFs are accurate and correct. If some assessments are not done, or if certain information is not available, not applicable or unknown, the Investigator shall indicate this in the eCRF. The Investigator shall electronically sign off the study data. By signing, the Investigator takes responsibility for the accuracy, completeness, and legibility of the data reported to the Sponsor in the eCRF.

2023-04-18 09:24

Doc id 43CH1627 Clinical Study Protocol GALDERMA MA-34970

#### 9.2.2 The query process

The monitor shall review the eCRFs and evaluate them for completeness and consistency by 100%. Each eCRF shall be compared with the respective source documents to ensure that there are no discrepancies between critical data. All entries, corrections, and alterations shall be made by the PI or his/her authorised designee. The monitor cannot enter data in the eCRFs. Once study data have been submitted to the central server via the eCRF, corrections to the data fields will be audit trailed, meaning that the reason for change, the name of the person who made the change, together with time and date will be logged. Roles and rights of the site personnel responsible for entering study data into the eCRF shall be determined in advance. If discrepant data is detected during review of the data, either by the Sponsor or its representatives, the responsible data manager or monitor shall raise a query in the electronic data capture application. The query shall state the question or data to be changed and shall be resolved in the system by the PI or his/her authorised designee. The appropriate study site personnel shall answer the queries in the eCRF. This will be audit trailed by the electronic data capture application meaning that the name of study site personnel, time, and date is logged.

#### 9.2.3 User identification

Electronic CRF records will be automatically appended with the identification of the creator, by means of their unique User ID. Specified records shall be electronically signed by the Investigator to document his/her review of the data and acknowledgement that the data are accurate. This will be facilitated by means of the Investigator's unique User ID and password; date and time stamps will be added automatically at time of electronic signature. If an entry in an eCRF requires change, the correction shall be made in accordance with the relevant software procedures.

#### 9.2.4 Audit trail

All changes will be fully recorded in a protected audit trail and a reason for the change shall be stated. Once all data have been entered, verified, and validated, the database will be locked.

#### 9.3 **Source documents**

The eCRF is essentially considered a data entry form and does not constitute the original (or source) medical records unless otherwise specified. Source documents are all documents used by the Investigator or hospital that relate to the subject's medical history, that verifies the existence of the subject, the inclusion and exclusion criteria, and all records covering the subject's participation in the study. They include photographs, memoranda, material dispensing records, subject files, etc.

The PI is responsible for maintaining source documents. These shall be made available for inspection by the monitor at each monitoring visit. The Investigator must submit a completed eCRF for each subject for whom signed informed consent has been collected. All supportive documentation submitted with the eCRF, such as photographs, should be clearly identified with the subject number. Any personal information, including name, shall be removed or rendered illegible to preserve individual confidentiality.



#### 9.4 Record keeping and access to source data

The PI/institution shall permit study-related monitoring, audits and IEC review and shall provide direct access to the source data/medical record including the identity of all participating subjects (sufficient information to link records, i.e. eCRF, medical records, original signed Informed Consent Forms and detailed records of study product accountability). The records should be retained by the PI as required by local legislation and international guidelines. Any transfer of responsibility for storage of the records shall be documented and the Sponsor should be informed in writing.

The Sponsor shall verify that each subject has consented in writing to direct access to the original medical record/source data (by the use of written subject information and signed informed consent). The data recorded in the eCRFs shall be checked for consistency with the source documents/medical record by the monitor during monitoring (source data verification; SDV). In order to be able to perform SDV, information about each subject's participation in the study has to be detailed in the medical record.

The source data location log specifies what data that should be available in the medical record. The source data location log should also specify the data for which the eCRF serves as the source. Such data only need to be recorded in the eCRF and are typically associated with study-specific procedures and not with normal clinical care practice. For this type of study data the Investigator would not be expected to duplicate the information into the medical record.

#### 9.5 Document and data retention

All records pertaining to the conduct of the study, including signed eCRFs, Informed Consent Forms, study product accountability records, source documents, and other study documentation must be retained after study completion according to national legislation and the CTA. Sponsor will inform the sites as to when these documents no longer needs to be retained. Measures should be taken to prevent accidental or premature destruction of these documents (e.g. protection against damage and unauthorised access, preferably by storage in a fire-proof cabinet). Refer to the CTA.

After study completion and database lock, a security sealed CD with electronic study data shall be provided by the eCRF vendor for archiving.

It is the PI's responsibility to inform Q-Med AB in writing if the Investigator file is moved or if the responsibility for the documents is transferred to someone else

#### 10 Statistical Methods

#### 10.1 General

A comprehensive Statistical Analysis Plan (SAP) with detailed description of all statistical analyses will be written and finalized prior to database lock (DBL). All statistical analyses, including summary tables and data listings, will be performed using the SAS® system (version 9.4 or later).

Print date:



Continuous variables will be summarised using standard statistical measures, such as mean, median, standard deviation, minimum and maximum values. Categorical variables will be presented in frequency tables with number and percent of observations for each level.

All confidence intervals will be two-sided and use the 95% confidence level. All statistical testing will be two-sided and performed at a significance level of 5%.

## 10.2 Analysis Populations

The following populations will be defined:

| • | Safety | Includes all subjects who were treated with Restylane Defyne or randomized to no-treatment group. Subjects are analyzed based on the as treated principle. |
|---|---|---|
| • | Full Analysis Set (FAS) | Includes all subjects who were treated with Restylane Defyne or randomized to no-treatment group. Subjects are analysed according to the randomisation assignment. |
| • | Per Protocol (PP) | Includes all subjects in FAS that comply to the protocol procedures with no deviations that can affect the evaluation of the primary variable. |

The FAS population is the primary population for all effectiveness analyses. All safety analyses will be based on the Safety population.

### 10.3 Demographics, baseline assessments, and subject characteristics

Demographic endpoints and subject characteristics will be presented by treatment group using descriptive statistics.

## 10.4 Effectiveness Analysis

#### Primary analysis

The percentage of responders (a responder will be defined as a subject with at least 1 point improvement from baseline GCRS) will be calculated for Restylane Defyne group at 6 months after last treatment, and for no treatment Control Group at 6 months after randomization based on the Blinded Evaluator's assessment.

In addition, for each group the two-sided 95% confidence intervals around the estimates of the percentage of responders will also be calculated.

# CC

#### Secondary analysis

The percentage of responders based on the GCRS will also be derived at all applicable follow-up visits for both the Blinded Evaluator's assessment and the Treating Investigator's

Effective date: 2018-01-15 10:39

43CH1627 Clinical Study Protocol

Doc id

Print date:

MA-34970

2023-04-18 09:24

assessment respectively. The response rates and their 95% confidence interval will be presented by visit and group.



## 10.5 Safety Analysis

CCI

A graph will be generated to illustrate the incidence over time. Number of days with the event will be summarized using mean, SD, min, max and median.

All AEs will be coded by preferred terms in the MedDRA dictionary.

Related AEs will be summarised by SOC, PT and intensity. In addition, for related AEs the number of days to onset and the duration of event will be summarised by SOC and PT and treatment using mean, SD, min, max and median.

Serious AEs will be listed.

Non-related AEs will be summarised by SOC, PT, and intensity and by treatment.

#### 10.6 Handling of Missing Data

Number of missing values will be summarized and reported as appropriate.

Different assumptions regarding the missing data will be used. For the primary effectiveness analysis, missing values in the FAS will be assumed to be missing due to lack of effect. Therefore missing data up to the Month 6 visit will be imputed using the baseline observation carried forward (BOCF) method. As an alternative approach, missing data will be assumed to be unrelated to treatment effect.

More details will be

given in the SAP. Both of these alternatives will estimate the effectiveness of the treatment policy (irrespective of use of unallowable treatments, procedures, or medications) rather than the true, clinical treatment effect.

To obtain an estimate of the true clinical treatment effect, the primary effectiveness analysis will be performed using the PP.

All other endpoints will be analysed on available data, i.e. no imputations will be done.

#### 10.7 Interim Analysis

An interim analysis is planned once all subjects in Treatment Group complete the 12 months visit after last treatment (or discontinued before) and all subjects in Control Group complete the 6 months visit after last treatment (or discontinued before).

#### 10.8 Data monitoring committee

Not applicable for this study.

#### 10.9 Withdrawals and deviations

All withdrawn subjects will be listed individually, including at least subject number, date and reason for withdrawal, and last visit performed.

Subjects with CSP deviations will be listed individually, including subject number and observed deviation. Depending on the seriousness of the deviation, subject might be excluded from the PP population, which shall be documented prior to DBL.

Deviations from the statistical plan will be documented in protocol Deviation log.

#### 10.10 Sample Size



account for 15% drop-outs, approximately 111 will be randomized to the Restylane Defyne Treatment Group and approximately 37 to the Control Group.

## 11 Protection of personal data

For the purposes of the study, Sponsor will be considered the data controller, and Institution and PI will both be considered data processors.

All processing of personal data must be carried out in accordance with national legislation concerning the protection of personal data. The Institution and the PI are responsible for complying with all requirements pursuant to national legislation in the country in which the Institution and the PI are located. The Sponsor will ensure that all requirements are complied with for data processing, which is carried out in Sweden by the Sponsor.

The Informed Consent Form shall contain information about what personal data to be collected in the study and that this will be kept confidential. The provided information shall be sufficient to enable all subjects to give their consent not only to the participation in the study, but also to the processing of personal data. Such information includes information regarding the purposes of the collecting, processing, data transfer to countries outside



Print date:

2023-04-18 09:24

China, and the length of time during which personal data will be stored. The subject shall have the right of access to stored personal data, and the right to correction of incorrect information. If a subject decides to terminate the study prematurely, data collected before withdraw of consent will be used in the evaluation of the study, however no new data may be collected. Authorised representatives from the Sponsor or a RA may visit the study site to perform audits/inspections, including source data verification, i.e. comparing data in the subjects' medical records and the eCRF. Data and information shall be handled strictly confidential.

## 12 Quality Control and Quality Assurance

### 12.1 Quality control

On-site monitoring of the study will be arranged by the Sponsor according to GCP guidelines to verify that the rights and well-being of the subjects are protected, the reported data are accurate, complete, verifiable from source documents, and that the conduct of the study complies with the approved CSP, subsequent amendment(s), GCP and the applicable regulatory requirements.

Any CSP deviation shall be reported in the eCRF, which shall be verified, discussed, and collected, by the monitor and appropriate corrective and preventive actions shall be taken. The PI is responsible for promptly reporting any deviations from the CSP that affects the rights, safety or well-being of the subject or the scientific integrity of the study, including those which occur under emergency circumstances, to the Sponsor as well as the IEC if required by national regulations. Deviations shall be reviewed to determine the need to amend the CSP or to terminate the study. Handling of CSP deviations shall be performed as described in the monitoring manual.

Prior to subject enrolment, all individuals involved in the conduct and/or surveillance of a clinical trial are made aware of the deviation categories and reporting requirements via information/training session ensured by the Clinical Trial Team.

## 12.2 Quality assurance

The study site may be subject to quality assurance audit by the Sponsor as well as inspection by appropriate RA. It is important that the PI and other relevant study site personnel are available during the monitoring visits, possible audits, and inspections, and that sufficient time is devoted to the monitoring process.

Each participating member of the study site team shall provide a curriculum vitae (CV) or equivalent that demonstrates their qualifications to conduct the study. The CV shall give name, date and place of birth, address and place of work, and shall show the training, appointments and, for the PI, any other information that confirms the suitability of the PI to be responsible for the study.

It is the responsibility of the PI to ensure that all personnel involved in the study are fully informed of all relevant aspects of the study, including detailed knowledge of and training in all procedures to be followed. All Investigators and other responsible persons shall be listed together with their function in the study on the signature and delegation log.

## 12.3 Changes to the clinical study protocol

The PI and other site personnel involved in the study must not implement any deviation from or changes to the CSP without agreement with the Sponsor and prior review and documented approval from the IEC, except where necessary to eliminate an immediate hazard to the subjects. All changes to the final CSP must be documented in a written protocol amendment. However, administrative changes are to be documented in the Sponsor file without requiring a protocol amendment.

## 13 Financing, Indemnification, and Insurance

The CTA outlines the compensation and payment terms of the study. The CTA must be signed before the first subject is screened in the study. If there are differences between the CTA and the CSP regarding certain rights and obligations, the CTA is the prevailing document. Q-Med AB's obligations in this clinical study are covered by Galderma's global general liability program. An insurance certificate will be provided upon request. The institution/PI is obligated to maintain insurance coverage for their obligations in the clinical study according to the CTA.

## 14 Publication Policy

The PI's, institutions, and Q-Med AB's obligations regarding intellectual property rights, confidentiality, and publications are described in detail in the CTA.

The aim is to submit the results of this study for publication in the public database ClinicalTrials.gov and to a medical journal for a first joint publication of the results. Everyone who is to be listed as an author of the results of this multicentre study shall have made a substantial, direct, intellectual contribution to the work. Authorship will be based on (1) substantial contributions to the conception or design of the work; or the acquisition, analysis, or interpretation of data for the work; and (2) drafting the work or revising it critically for important intellectual content; and (3) final approval of the version to be published; and (4) agreement to be accountable for all aspects of the work in ensuring that questions related to the accuracy or integrity of any part of the work are appropriately investigated and resolved\*. Conditions 1, 2, 3, and 4 must all be met in order to be designated as author. Those who do not meet all four criteria should be acknowledged. Among the authors that fulfil the above mentioned criteria, one author will be appointed by Q-Med AB to take primary responsibility for the overall work as primary author.

\*Defining the role of authors and contributors, compiled by the International Committee of Medical Journal Editors (ICMJE) (http://www.icmje.org).

# 15 Suspension or Premature Termination

The Sponsor will suspend or terminate the study when so instructed by the IEC or if it is judged that the subjects are subjected to unreasonable risks, or for valid scientific or administrative reasons.

Print date:

2023-04-18 09:24

The Sponsor may also decide to close a single study site due to unsatisfactory subject enrolment or non-compliance with the CSP, GCP, or applicable regulatory requirements.

In the event of premature termination, Q-Med AB will provide information on the handling of currently enrolled subjects who have not completed the study

Doc id 43CH1627 Clinical Study Protocol GALDERMA MA-34970

Print date:

2023-04-18 09:24

### 16 References

- Monheit GD, Coleman KM. Hyaluronic acid fillers. Dermatol 2006 May-Jun; 19(3):141-50.
- Gold M. The science and art of hyaluronic acid dermal filler use in esthetic applications. J Cosmet Dermatol 2009 Dec; 8(4):301-7.
- Pons-Guiraud A. Classification des produits de comblement disponsible en France. Ann Dermatol Venerol 2008;135:I S27-34.
- Ascher B et al. Chapter 34: Hyaluronic acids. In: Ascher B ed. Injection Treatment in Cosmetic Surgery. Informa UK Ltd. 2009.
- Talarico S et al. High Patient Satisfaction of a Hyaluronic Acid Filler Producing Enduring Full-Facial Volume Restoration: An 18-Month Open Multicenter Study. Dermatologic Surgery 2015, 41(12):1361-1369.
- Rzany,B., et al. Full-face rejuvenation using a range of hyaluronic acid fillers: efficacy, safety, and patient satisfaction over 6 months. Dermatol. Surg 2012a. 38, 1153-1161.
- Kestemont, P et al. Sustained efficacy and high patient satisfaction after cheek enhancement with a new hyaluronic acid dermal filler. J Drugs Dermatol 2012. 11, s9-16.
- Farhi, D., et al. The Emervel French survey: a prospective real-practice descriptive study of 1,822 patients treated for facial rejuvenation with a new hyaluronic acid filler. J Drugs Dermatol 2013; 12, e88-e93.
- Galderma Chin Retrusion Scale Validation Report (internal document MA-33370).
- 10. Weiss RA et al. Effectiveness and Safety of Large Gel Particle Hyaluronic Acid with Lidocaine for Correction of Midface Volume Deficit or Contour Deficiency. Dermatol Surg. 2016 Jun; 42(6):699-709.
- 11. Glogau RG et al. A randomized, evaluator-blinded, controlled study of the effectiveness and safety of small gel particle hyaluronic acid for lip augmentation. Dermatol Surg. 2012 Jul;38(7 Pt 2):1180-92.
- 12. Galderma. A pivotal USA randomized evaluator-blinded, active-controlled, multi-center, splitface comparison study of Emervel® Deep Lidocaine versus Juvederm® Ultra Plus in the treatment of moderate to severe facial wrinkles and folds. Clinical Investigationa Report: RD.06.CIR.18156. 2013.
- 13. Galderma. A phase IV European randomized, evaluator-blinded, controlled, multi-center, intraindividual right-left comparison study of Evenor Deep versus Perlane in the treatment of soft tissue contour deformities. Clinical Investigational Report: RD.03.SRE.40072. 2011.
- 14. Ascher B, et al. Efficacy and safety of a new hyaluronic acid dermal filler in the treatment of severe nasolabial lines - 6-month interim results of a randomized, evaluator-blinded, intra-individual comparison study . J Cosmet Dermatol. 2011 Jun;10(2):94-8.
- 15. Rzany B, Cartier H, Kestermont P, Trevidic P, Sattler G, Kerrouche N, Dhuin JC. Correction of tear troughs and periorbital lines with a range of customized hyaluronic acid fillers. J Drugs Dermatol. 2012 Jan;11(1 Suppl):s27-34.
- 16. Cartier H, Trevidic P, Rzany B, Sattler G, Kestemont P, Kerrouche N, Dhuin JC. Perioral rejuvenation with a range of customized hyaluronic acid fillers: efficacy and safety over six months with a specific focus on the lips. J Drugs Dermatol. 2012 Jan;11(1 Suppl):s17-26.
- 17. Talarico S, et al. High Patient Satisfaction of a Hyaluronic Acid Filler Producing Enduring Full-Facial Volume Restoration: An 18-Month Open Multicenter Study. Dermatol Surg. 2015 Dec;41(12):1361-9.
- 18. Zhou J, et al. Chin augmentation with hyaluronic acid injection. Chin J Aesth Plast Surg. 2014 Jan; 11 (1): 26-28.
- 19. Zhang HJ, et al. Clinical application and observation of injectable modified sodium hyaluronate gel filler for facial cosmetic surgery. Zhonghua Kou Qiang Yi Xue Za Zhi. 2017 Mar 9;52(3):194-197.

43CH1627 Clinical Study Protocol Doc id 👶 GALDERMA MA-34970

# 17 Appendices

Appendix 1 Declaration of Helsinki

Appendix 2 Photo guide for Galderma Chin Retrusion Scale

GALDERMA

Title

43CH1627 Clinical Study Protocol

MA-34970

Appendix 1

Declaration of Helsinki

Print date:

2023-04-18 09:24

# WMA Declaration of Helsinki - Ethical Principles for Medical Research Involving Human Subjects

Adopted by the 18th WMA General Assembly, Helsinki, Finland, June 1964 and amended by the:

29th WMA General Assembly, Tokyo, Japan, October 1975

35th WMA General Assembly, Venice, Italy, October 1983

41st WMA General Assembly, Hong Kong, September 1989

48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996

52nd WMA General Assembly, Edinburgh, Scotland, October 2000

53rd WMA General Assembly, Washington DC, USA, October 2002 (Note of Clarification added)

55th WMA General Assembly, Tokyo, Japan, October 2004 (Note of Clarification added)

59th WMA General Assembly, Seoul, Republic of Korea, October 2008

64th WMA General Assembly, Fortaleza, Brazil, October 2013

#### **Preamble**

1. The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving human subjects, including research on identifiable human material and data.

The Declaration is intended to be read as a whole and each of its constituent paragraphs should be applied with consideration of all other relevant paragraphs.

Consistent with the mandate of the WMA, the Declaration is addressed primarily to physicians. The WMA encourages others who are involved in medical research involving human subjects to adopt these principles.

#### **General Principles**

- 3. The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 4. It is the duty of the physician to promote and safeguard the health, well-being and rights of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfilment of this duty.
- 5. Medical progress is based on research that ultimately must include studies involving human subjects.
- 6. The primary purpose of medical research involving human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the best proven interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.
- 7. Medical research is subject to ethical standards that promote and ensure respect for all human subjects and protect their health and rights.
- 8. While the primary purpose of medical research is to generate new knowledge, this goal can never take precedence over the rights and interests of individual research subjects.
- 9. It is the duty of physicians who are involved in medical research to protect the life, health, dignity, integrity, right to self-determination, privacy, and confidentiality of personal information of research subjects. The responsibility for the protection of research subjects must always rest with the physician

# Declaration of Helsinki

Print date:

2023-04-18 09:24

or other health care professionals and never with the research subjects, even though they have given consent.

- 10. Physicians must consider the ethical, legal and regulatory norms and standards for research involving human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research subjects set forth in this Declaration.
- 11. Medical research should be conducted in a manner that minimises possible harm to the environment.
- 12. Medical research involving human subjects must be conducted only by individuals with the appropriate ethics and scientific education, training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional.
- 13. Groups that are underrepresented in medical research should be provided appropriate access to participation in research.
- 14. Physicians who combine medical research with medical care should involve their patients in research only to the extent that this is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research study will not adversely affect the health of the patients who serve as research subjects.
- 15. Appropriate compensation and treatment for subjects who are harmed as a result of participating in research must be ensured.

#### Risks, Burdens and Benefits

- 16. In medical practice and in medical research, most interventions involve risks and burdens. Medical research involving human subjects may only be conducted if the importance of the objective outweighs the risks and burdens to the research subjects.
- 17. All medical research involving human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and groups involved in the research in comparison with foreseeable benefits to them and to other individuals or groups affected by the condition under investigation.
  - Measures to minimise the risks must be implemented. The risks must be continuously monitored, assessed and documented by the researcher.
- 18. Physicians may not be involved in a research study involving human subjects unless they are confident that the risks have been adequately assessed and can be satisfactorily managed.
  - When the risks are found to outweigh the potential benefits or when there is conclusive proof of definitive outcomes, physicians must assess whether to continue, modify or immediately stop the study.

#### **Vulnerable Groups and Individuals**

- 19. Some groups and individuals are particularly vulnerable and may have an increased likelihood of being wronged or of incurring additional harm.
  - All vulnerable groups and individuals should receive specifically considered protection.
- 20. Medical research with a vulnerable group is only justified if the research is responsive to the health needs or priorities of this group and the research cannot be carried out in a non-vulnerable group. In

Declaration of Helsinki

Print date:

2023-04-18 09:24

addition, this group should stand to benefit from the knowledge, practices or interventions that result from the research.

#### **Scientific Requirements and Research Protocols**

- 21. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- 22. The design and performance of each research study involving human subjects must be clearly described and justified in a research protocol.

The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, sponsors, institutional affiliations, potential conflicts of interest, incentives for subjects and information regarding provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the research study.

In clinical trials, the protocol must also describe appropriate arrangements for post-trial provisions.

#### **Research Ethics Committees**

23. The research protocol must be submitted for consideration, comment, guidance and approval to the concerned research ethics committee before the study begins. This committee must be transparent in its functioning, must be independent of the researcher, the sponsor and any other undue influence and must be duly qualified. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research subjects set forth in this Declaration.

The committee must have the right to monitor ongoing studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No amendment to the protocol may be made without consideration and approval by the committee. After the end of the study, the researchers must submit a final report to the committee containing a summary of the study's findings and conclusions.

#### **Privacy and Confidentiality**

24. Every precaution must be taken to protect the privacy of research subjects and the confidentiality of their personal information.

#### **Informed Consent**

- 25. Participation by individuals capable of giving informed consent as subjects in medical research must be voluntary. Although it may be appropriate to consult family members or community leaders, no individual capable of giving informed consent may be enrolled in a research study unless he or she freely agrees.
- 26. In medical research involving human subjects capable of giving informed consent, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail, post-study provisions and any other relevant aspects of the study. The potential subject must be informed of the right to refuse to participate in the study or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential subjects as well as to the methods used to deliver the information.

# Declaration of Helsinki

Print date:

2023-04-18 09:24

After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.

All medical research subjects should be given the option of being informed about the general outcome and results of the study.

- 27. When seeking informed consent for participation in a research study the physician must be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent must be sought by an appropriately qualified individual who is completely independent of this relationship.
- 28. For a potential research subject who is incapable of giving informed consent, the physician must seek informed consent from the legally authorised representative. These individuals must not be included in a research study that has no likelihood of benefit for them unless it is intended to promote the health of the group represented by the potential subject, the research cannot instead be performed with persons capable of providing informed consent, and the research entails only minimal risk and minimal burden.
- 29. When a potential research subject who is deemed incapable of giving informed consent is able to give assent to decisions about participation in research, the physician must seek that assent in addition to the consent of the legally authorised representative. The potential subject's dissent should be respected.
- 30. Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research group. In such circumstances the physician must seek informed consent from the legally authorised representative. If no such representative is available and if the research cannot be delayed, the study may proceed without informed consent provided that the specific reasons for involving subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research must be obtained as soon as possible from the subject or a legally authorised representative.
- 31. The physician must fully inform the patient which aspects of their care are related to the research. The refusal of a patient to participate in a study or the patient's decision to withdraw from the study must never adversely affect the patient-physician relationship.
- 32. For medical research using identifiable human material or data, such as research on material or data contained in biobanks or similar repositories, physicians must seek informed consent for its collection, storage and/or reuse. There may be exceptional situations where consent would be impossible or impracticable to obtain for such research. In such situations the research may be done only after consideration and approval of a research ethics committee.

#### **Use of Placebo**

33. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best proven intervention(s), except in the following circumstances:

Where no proven intervention exists, the use of placebo, or no intervention, is acceptable; or

Where for compelling and scientifically sound methodological reasons the use of any intervention less effective than the best proven one, the use of placebo, or no intervention is necessary to determine the efficacy or safety of an intervention

# Declaration of Helsinki

Print date:

2023-04-18 09:24

and the patients who receive any intervention less effective than the best proven one, placebo, or no intervention will not be subject to additional risks of serious or irreversible harm as a result of not receiving the best proven intervention.

Extreme care must be taken to avoid abuse of this option.

#### **Post-Trial Provisions**

34. In advance of a clinical trial, sponsors, researchers and host country governments should make provisions for post-trial access for all participants who still need an intervention identified as beneficial in the trial. This information must also be disclosed to participants during the informed consent process.

#### **Research Registration and Publication and Dissemination of Results**

- 35. Every research study involving human subjects must be registered in a publicly accessible database before recruitment of the first subject.
- 36. Researchers, authors, sponsors, editors and publishers all have ethical obligations with regard to the publication and dissemination of the results of research. Researchers have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. All parties should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results must be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest must be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

#### **Unproven Interventions in Clinical Practice**

37. In the treatment of an individual patient, where proven interventions do not exist or other known interventions have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorised representative, may use an unproven intervention if in the physician's judgement it offers hope of saving life, re-establishing health or alleviating suffering. This intervention should subsequently be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information must be recorded and, where appropriate, made publicly available.

Print date: 2023-04-18 09:24

GALDERMA

Title

43CH1627 Clinical Study Protocol

MA-34970

Appendix 2
Photo guide for GCRS

# **Galderma Chin Retrusion Scale**



Version: 3.0 Effective date: 2018-01-15 10:39

GALDERMA

Title
43CH1627 Clinical Study Protocol

MA-34970

Appendix 3

Print date:

2023-04-18 09:24



Print date: 2023-04-18 09:24 43CH1627 Clinical Study Protocol Doc id ♣ GALDERMA MA-34970 Appendix 3

# SIGNATURES PAGE

| Date | Signed by |
|------------------|------------------------------|
| 2018-01-15 07:26 | PPD |
| Justification | Approved by Technical Expert |
| 2018-01-15 07:30 | PPD |
| Justification | Approved by Project Manager |
| 2018-01-15 08:33 | PPD |
| Justification | Approved by Technical Expert |
| 2018-01-15 10:39 | PPD |
| Justification | Approved by Owner |